25 August 2025

| Protocol:<br>NCT No.:<br>Subject: | NKF-INS(A)-101<br>06492226<br>Cover Letter for Protocol |
|---|---|
| Protocol V2.0 06MAY202 | 24 for NKF-INS(A)-101 is attached with NCT06492226. |
| Sincerely, | |
| Chris Schroth<br>Clinical Project Manager | Xentria, Inc. |

#### CLINICAL STUDY PROTOCOL



Xentria, Inc.

Protocol Title: A single-center, single-dose, double-blind, randomized, three-period, three-treatment, six-sequence, crossover study to demonstrate pharmacokinetic and pharmacodynamic similarity between NKF-INS(A), US-NovoLog®, and EU-NovoRapid® using the euglycemic clamp technique in healthy male adult volunteers

Protocol Number: NKF-INS(A)-101

**IND Number:** 170945

EU Clinical Trial Number: Not applicable

Name of Investigational Product: NKF-INS(A) (Proposed Biosimilar to Insulin Aspart)

**Phase of Development:** Phase 1

**Indication:** Diabetes Mellitus

**Sponsor:** Xentria, Inc.

2071 N. Southport Ave. Chicago, IL 60614 USA Tel: 224-443-4615

Email: contact@xentria.com

Protocol Version: 2.0

**Protocol Date:** 06-May-2024

#### -CONFIDENTIAL-

This document is a confidential communication of Xentria, Inc. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Xentria, Inc. except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered. Furthermore, the information is only meant for review and compliance by the recipient, his or her staff, and applicable institutional review committee and regulatory agencies to enable conduct of the study.

**Sponsor Signatories:** 

#### PROTOCOL APPROVAL SIGNATURES

| Protocol Title: | A single-center, single-dose, double-blind, randomized, three-period, |
|---|---|
| | three-treatment, six-sequence, crossover study to demonstrate |
| | pharmacokinetic and pharmacodynamic similarity between NKF-INS(A), |
| | US-NovoLog®, and EU-NovoRapid® using the euglycemic clamp technique |
| | in healthy male adult volunteers |
| Protocol Number: | NKF-INS(A)-101 |

This study will be conducted in full conformance with the International Council for Harmonisation (ICH) E6 (R2) guideline for Good Clinical Practice (GCP) and the principles of the Declaration of Helsinki, or all relevant laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the European Union (EU) or European Economic Area will comply with the EU Clinical Trial Regulation (EU-CTR).

| Tom Matthews | |
|--------------------------------------|--------------------|
| Vice President, Clinical Development | <u></u> |
| Xentria, Inc. | Signature and Date |

#### INVESTIGATOR SIGNATURE PAGE

**Protocol Title:** A single-center, single-dose, double-blind, randomized, three-period, three-treatment,

six-sequence, crossover study to demonstrate pharmacokinetic and pharmacodynamic similarity between NKF-INS(A), US-NovoLog®, and EU-NovoRapid® using the

euglycemic clamp technique in healthy male adult volunteers

**Protocol Number:** NKF-INS(A)-101

This study will be conducted in full conformance with the International Council for Harmonisation (ICH) E6 (R2) guideline for Good Clinical Practice (GCP) and the principles of the Declaration of Helsinki, or all relevant laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the European Union (EU) or European Economic Area will comply with the EU Clinical Trial Regulation (EU-CTR).

- I, the undersigned, have reviewed this protocol including appendices, and I will conduct the study as described in compliance with this protocol, GCP, and relevant ICH guidelines.
- I am thoroughly familiar with the appropriate use of the study treatment, as described in this protocol and
  any other information provided by Xentria, Inc. including, but not limited to, the current Investigator's
  Brochure.
- After the protocol has been approved by the Independent Ethics Committee (IEC)/Institutional Review
  Board (IRB), I will not modify this protocol. I will submit the protocol amendments and/or any informed
  consent form modifications to Xentria, Inc. and the IEC/IRB, and approval will be obtained before any
  amendments are implemented.
- I ensure that all persons or parties assisting me with the study are adequately qualified, trained, and informed about the Xentria, Inc. study treatment and of their delegated study-related duties and functions as described in the protocol.
- I ensure that source documents and study records that include all pertinent observations on each of the site's study participants are attributable, legible, contemporaneous, original, accurate, and complete, consistent, enduring, and available.
- I understand that all information obtained during the conduct of the study with regard to the participants' state of health will be regarded as confidential. No participants' personal identifying information will be disclosed. All participants will be identified by assigned numbers on all case report forms, laboratory samples, or source documents forwarded to the Sponsor. Clinical information may be reviewed by the Sponsor or its agents or regulatory agencies. Agreement must be obtained from the participant before disclosure of participant information to a third party.
- Information developed in this clinical study may be disclosed by Xentria, Inc. to other clinical Investigators, regulatory agencies, or other health authority or government agencies as required.

| Name: | |
|--------------|------------------------|
| Title: | Investigator Signature |
| Institution: | |
| | Date (DD-MMM-YYYY) |

## 1. SYNOPSIS

| Title of Study | six-sequence, crossover similarity between NKF- | ose, double-blind, randomized, three-period, three-treatment, study to demonstrate pharmacokinetic and pharmacodynamic INS(A), US-NovoLog <sup>®</sup> , and EU-NovoRapid <sup>®</sup> using the ique in healthy male adult volunteers |
|---|---|---|
| <b>Protocol Number</b> | NKF-INS(A)-101 | |
| Investigators/Stud<br>Sites | y This is a single-center str | udy that will be conducted in South Africa |
| Phase of<br>Development | Phase 1 | |
| Purpose and Rationale | Despite advances in diab<br>cost-effective insulins in | etes mellitus care, there remains a critical unmet need for many markets. |
| | hypoglycemia, are exper<br>NovoLog® in the United<br>has a faster onset and a s<br>control by means of lowe<br>As a biosimilar to insulin<br>medical need in patients<br>NKF-INS(A) to EU-Nov | time insulin analogues, while associated with a lower risk of asive. Insulin aspart is a rapid-acting insulin marketed as States (US) and NovoRapid® in the European Union (EU). It horter duration of action, resulting in postprandial glycemic ering the total glucose excursion following a meal. In aspart, NKF-INS(A) has the potential to address this unmet with diabetes mellitus. In order to demonstrate biosimilarity of roRapid® and US-NovoLog®, a Phase 1 study will evaluate the (A) to the reference products using a euglycemic clamp e volunteers. |
| Objectives | | Endpoints |
| Primary | | |
| <ul> <li>To compare th<br/>US-approved a<br/>aspart to demo<br/>insulin aspart.</li> <li>To compare th<br/>US-approved a</li> </ul> | e PK of NKF-INS(A) to nd EU-authorized insulin nstrate PK similarity for e PD of NKF-INS(A) to nd EU-authorized insulin by examining GIR profiles C dose. | <ul> <li>Aspart concentration-time curve from 0 to 12 hours (AUC<sub>0-t</sub>)</li> <li>Maximum observed insulin aspart concentration (C<sub>max</sub>)</li> <li>Area under the GIR-time curve from 0 to 12 hours (AUCGIR<sub>0-t</sub>)</li> <li>Maximum GIR (GIR<sub>max</sub>) of glucose.</li> </ul> |
| <ul> <li>To compare the US-approved a aspart to demo insulin aspart.</li> <li>To compare the US-approved a aspart injection</li> </ul> | nd EU-authorized insulin<br>nstrate PK similarity for<br>e PD of NKF-INS(A) to<br>nd EU-authorized insulin<br>by examining GIR profiles | <ul> <li>(AUC<sub>0-t</sub>)</li> <li>Maximum observed insulin aspart concentration (C<sub>max</sub>)</li> <li>Area under the GIR-time curve from 0 to 12 hours (AUCGIR<sub>0-t</sub>)</li> </ul> |

| action (duration of action) |
|---|
| AE assessments (including injection site reactions),<br>clinical laboratory investigations (hematology, clinical<br>chemistry [including glucose], coagulation, and<br>urinalysis), vital signs, physical examinations, 12-lead<br>ECG, prior and concomitant medication assessments |
| <ul> <li>Corrected and uncorrected C-peptide concentrations</li> <li>If possible, i.e., if the terminal phase of serum concentration-time profile has sufficient data points, apparent terminal elimination half-life (t½.z), apparent terminal elimination rate constant (λz), mean residence time (MRT), clearance (CL/F), and volume of distribution (V/F) will be calculated</li> </ul> |
| d |

#### **Study Design**

Study NKF-INS(A)-101 is a Phase 1, 12-hour euglycemic glucose clamp study conducted using a randomized, double-blind, three-period, three-treatment, six-sequence, crossover design. The study will compare single doses of the proposed insulin biosimilar (NKF-INS(A)) with respective EU- and US-reference products in healthy male participants.

Written informed consent will be obtained from all participants, and the study will be conducted in accordance with the principles of Good Clinical Practice (GCP) as defined by the International Conference of Harmonization (ICH).

The study will consist of several visits: a screening visit to obtain informed consent and assess eligibility for participation, three dosing visits with a washout period between each visit, and a follow-up visit after the last dose.

Three insulin products (NKF-INS(A), EU-NovoRapid<sup>®</sup>, and US-NovoLog<sup>®</sup>) will be administered over three treatment periods. Upon admission to the clinical research unit (CRU) on Day -1, participants will be randomized to one of six treatment sequences in a 1:1:1:1:1 ratio, receiving a single subcutaneous (SC) dose of 0.3 U/kg administration of one of the three study drugs on each dosing day.

A 12-hour euglycemic glucose clamp will be conducted using a manual clamp technique, which will monitor the subject's blood glucose and administer glucose infusion (GIR) to maintain blood glucose close to the target blood glucose concentration. The clamp procedure will be initiated, maintained, and terminated, in accordance with the site standard operating procedures (SOPs). The participant's blood glucose will be maintained within a pre-defined target window per site SOP and clinical judgment for the participant by manually adjusting the GIR.

Blood samples will be collected at pre-specified intervals before and up to 12 hours after dosing for measurement of blood glucose, serum insulin, and C-peptide.

## Selection of Participants

#### **Inclusion Criteria**

Individuals must meet all of the following inclusion criteria to be included in the study:

- 1. Signed and dated informed consent obtained before any trial-related activities.

  Trial-related activities are any procedures that would not have been done during normal management of the participant
- 2. Healthy male participants
- 3. Age between 18 and 50 years, both inclusive
- 4. Body Mass Index between 18.5 and 29.0 kg/m<sup>2</sup>, both inclusive
- 5. Body weight  $\geq$  50 kg
- 6. Fasting plasma glucose concentration  $\leq$  5.5 mmol/L at screening
- 7. Considered generally healthy upon completion of medical history, physical examination, vital signs, electrocardiogram (ECG), and analysis of laboratory safety variables, as judged by the Investigator
- 8. Willing and able to comply with scheduled visits, treatment plan, clinical laboratory tests, and other study procedures including lifestyle considerations.
- 9. Participants must agree to use condoms during sexual intercourse. Additionally, female partners of male participants should use highly effective contraception. All contraceptive measures apply from screening until 90 days after study

| days after administration of study treatment. 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergie reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of su acute infection with fever or infectious disease | Reference Therapy | EU-NovoRapid® and US-NovoLog®, both administered as a 0.3 U/kg single SC dose in the periumbilical area. |
|---|---|---|
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergie reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergie reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dl. 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14. Have positive test results for hepatitis B surface antigen (HBsAg), immunoglobulim M (IgM) antibody t | | EUND:-IRI IC NIR 14I ' ' ' I O 2 IIII ' I CC I ' |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of macute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14. | _ | NKF-INS(A) administered as a 0.3 U/kg single SC dose in the periumbilical area. |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14. H | Size | 36 evaluable participants. |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening. 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level =140.4 mg/dl. 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14. Have positive test results for hepatitis B surface antigen (HBsAg), immunoglobulin M (IgM) antibody | Planned Sample | 54 healthy male participants are planned to be enrolled in the study to have at least |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥ 140.4 my/dl. 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14. | | |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria:</li> <li>1. Positive for human insulin antibodies at Screening</li> <li>2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> <li>3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.</li> <li>5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study drug; or of interfering with the interpretation of data.</li> <li>7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.</li> <li>8. Clinically significant abnormal ECG at screening.</li> <li>9. Glycemia level ≥140.4 mg/dl. 2 hours after the glucose load.</li> <li>10. Show evidence of significant active neuropsychiatric disease.</li> <li>11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year.</li> <li>12. Show evidence of human inmunodeficiency virus (HIV) infection and/or positive human HIV antibod</li></ul> | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening. 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or climination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dl. 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14 | | <u> </u> |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level 2140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14. | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergie reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. 14. | | medication within 14 days prior to dosing (apart from vitamin/mineral |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. 13. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergie reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergie reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening. | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load. 10. Show evidence of significant active neuropsychiatric disease. 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year. 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment. | | |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria: <ol> <li>Positive for human insulin antibodies at Screening</li> <li>Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.</li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.</li> <li>Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.</li> <li>Clinically significant abnormal ECG at screening.</li> <li>Glycemia level ≥140.4 mg/dL 2 hours after the glucose load.</li> <li>Show evidence of significant active neuropsychiatric disease.</li> <li>Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year.</li> </ol></li></ul> <li>Show evidence of an acute infection with fever or infectious disease at the time</li> | | 13. Show evidence of human immunodeficiency virus (HIV) infection and/or |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria: <ol> <li>Positive for human insulin antibodies at Screening</li> <li>Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.</li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.</li> <li>Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.</li> <li>Clinically significant abnormal ECG at screening.</li> <li>Glycemia level ≥140.4 mg/dL 2 hours after the glucose load.</li> <li>Show evidence of significant active neuropsychiatric disease.</li> <li>Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year.</li> </ol></li></ul> | | |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria:</li> <li>1. Positive for human insulin antibodies at Screening</li> <li>2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> <li>3. Have known allergics to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.</li> <li>5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.</li> <li>7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.</li> <li>8. Clinically significant abnormal ECG at screening.</li> <li>9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load.</li> <li>10. Show evidence of significant active neuropsychiatric disease.</li> <li>11. Positive urine drug test at screening and/or evidence of current use of known</li> </ul> | | |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria:</li> <li>1. Positive for human insulin antibodies at Screening</li> <li>2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> <li>3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.</li> <li>5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.</li> <li>7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.</li> <li>8. Clinically significant abnormal ECG at screening.</li> <li>9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load.</li> </ul> | | 11. Positive urine drug test at screening and/or evidence of current use of known |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator. 8. Clinically significant abnormal ECG at screening. | | 1 |
| <ol> <li>Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria: <ol> <li>Positive for human insulin antibodies at Screening</li> <li>Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> </ol> </li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.</li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.</li> <li>Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.</li> </ol> | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data. | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or | | interfering with the interpretation of data. |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological | | |
| <ol> <li>Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria: <ol> <li>Positive for human insulin antibodies at Screening</li> <li>Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> </ol> </li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.</li> <li>Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.</li> <li>Have clinically relevant history of or current cardiovascular, respiratory,</li> </ol> | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. 5. Have known allergies to insulin, its excipients, or related drugs or have history | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes. | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any | | |
| 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria Individuals will be excluded from participation if they meet any of the following criteria: 1. Positive for human insulin antibodies at Screening 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study. 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin. | | |
| <ol> <li>Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria: <ol> <li>Positive for human insulin antibodies at Screening</li> </ol> </li> <li>Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.</li> </ol> | | of relevant allergic reactions of any origin. |
| <ol> <li>Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria: <ol> <li>Positive for human insulin antibodies at Screening</li> </ol> </li> <li>Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be</li> </ol> | | |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria:</li> <li>1. Positive for human insulin antibodies at Screening</li> <li>2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives</li> </ul> | | enrolled in any other type of medical research study and judged not to be |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria:</li> <li>1. Positive for human insulin antibodies at Screening</li> </ul> | | |
| <ul> <li>10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.</li> <li>Exclusion Criteria</li> <li>Individuals will be excluded from participation if they meet any of the following criteria:</li> </ul> | | |
| Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted. Exclusion Criteria | | |
| 10. Have competence in speaking, writing, and comprehending the local | | Exclusion Criteria |
| days atten administration of study treatment | | |
| treatment male participants must refrain from donating or banking sperm for 90 | | |

| Treatment Duration Pharmacokinetics Pharmacodynamics | The study will consist of a screening period of up to 4 weeks (Days -28 to -1), three treatment periods each consisting of 1-day dose administrations and euglycemic clamp periods (periods 1, 2, and 3) separated by a washout period of 3-14 calendar days between treatment periods 1 and 2, and a washout period of 5-21 calendar days between treatment periods 2 and 3, and a follow-up period of 2-11 days. The entire study duration will be a maximum of 11 weeks. Insulin (serum) samples will be collected at 60, 30, 0 minutes pre-dose and 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 135, 150, 180, 210, 240, 300, 600, and 720 minutes post-dose. C-peptide (serum) 60, 30, 0 minutes pre-dose and 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 135, 150, 180, 210, 240, 300, 600, and 720 minutes post-dose. Blood glucose values will be analyzed pre-dose, every 3 minutes from 0 to 120 minutes, every 5 from 120 to 240 minutes, and every 10 minutes from 240 to 720 minutes post-dose. |
|---|---|
| Immunogenicity | Not applicable |
| Other Assessments | Safety assessments include vital signs, physical examinations, ECG recordings, clinical laboratory assessments (hematology, clinical chemistry [including glucose], coagulation, and urinalysis), AE monitoring (including injection site reactions). AEs will be coded by using the Medical Dictionary for Regulatory Activities dictionary. All treatment-emergent AEs (TEAEs) will be summarized by insulin product (NKF-INS(A), US-NovoLog®, EU-NovoRapid®) as follows: • All AEs • Grade ≥3 AEs • AEs related to study treatment, including related Grade ≥3 AEs • All adverse reactions • Serious AEs (SAEs) All AE data will be defined in the listing (onset, stop date, severity, etc.). The original results and change from baseline values for clinical laboratory assessments, vital signs, and ECG parameters, will be summarized by insulin product and scheduled visits. Potential clinically significant values will also be flagged and summarized. Significant changes in physical examination findings will be listed as AEs. Injection site reactions will be summarized by treatment group and scheduled visits. The number and percentage of participants having reactions at each assessment timepoint, overall and by specific reaction subtype, will be presented. Not applicable |
| Statistical Methods<br>and Planned<br>Analyses | The statistical evaluation will be performed using R version 4.0 or higher. All data will be listed, and summary tables and figures will be provided. Summary statistics will be presented by treatment group, to the extent possible. For continuous variables, data will be summarized with the number of participants (N), arithmetic mean, standard deviation (SD), median, minimum, and maximum by treatment group. Geometric mean and coefficient of variation (CV%) will be presented as appropriate, by treatment group. For categorical variables, data will be tabulated with the number and proportion of participants for each category by treatment group. |
| Interim Analysis | Not applicable. |

| Data Monitoring | Not applicable. |
|-----------------|-----------------|
| Committee | |

## 2. TABLE OF CONTENTS

| CLINIC | AL STUDY PROTOCOL | 1 |
|---|---|---|
| 1. | SYNOPSIS | 4 |
| 2. | TABLE OF CONTENTS | 10 |
| 3. | LIST OF ABBREVIATIONS | 15 |
| 4. | INTRODUCTION | 17 |
| 4.1. | Background on NKF-INS(A) | 17 |
| 4.1.1. | Preliminary Analytical Similarity Study for Program Feasibility | 17 |
| 4.2. | Clinical Benefits/Risks of NKF-INS(A) | 18 |
| 4.3. | Study Rationale | 18 |
| 4.4. | Dose Rationale | 18 |
| 5. | STUDY OBJECTIVES AND ENDPOINTS | 19 |
| 6. | INVESTIGATIONAL PLAN | 21 |
| 6.1. | Description of Overall Study Design and Plan | 21 |
| 6.2. | Discussion of Study Design | 22 |
| 6.3. | End of Study | 23 |
| 6.4. | Criteria for Early Study Termination | 23 |
| 7. | SELECTION OF STUDY POPULATION | 24 |
| 7.1. | Inclusion Criteria | 24 |
| 7.2. | Exclusion Criteria | 24 |
| 7.3. | Rescreening. | 25 |
| 7.4. | Study Withdrawal, Removal, and Replacement of Participants | 26 |
| 7.4.1. | Replacement of Participants | 26 |
| 8. | TREATMENTS | 27 |
| 8.1. | Study Treatment Description | 27 |
| 8.1.1. | Preparation, Handling, and Disposal | 28 |
| 8.1.2. | Product Labeling and Packaging | 28 |
| 8.1.3. | Administration | 28 |
| 8.1.4. | Storage | 28 |
| 8.2. | Dosage Schedule | 29 |
| 8.3. | Measures to Minimize Bias: Study Treatment Assignment and Blinding | 29 |
| 8.3.1. | Method of Study Treatment Assignment | 29 |

| 8.3.2. | Blinding | 29 |
|---|---|---|
| 8.4. | Treatment Modifications and Discontinuations | 30 |
| 8.5. | Treatment Accountability and Compliance | 31 |
| 8.6. | Prior and Concomitant Therapy and Other Restrictions During the Study | 31 |
| 8.6.1. | Prior and Concomitant Medications | 31 |
| 8.6.1.1. | Permitted Concomitant Medications and Therapies | 32 |
| 8.6.1.2. | Prohibited Concomitant Medications and Therapies | |
| 8.6.1.3. | Advisory on COVID-19 Vaccination and Risk Assessment | 32 |
| 8.6.2. | Other Restrictions During the Study | 33 |
| 8.6.2.1. | Meals and Dietary Restrictions | 33 |
| 8.6.2.2. | Caffeine, Alcohol and Tobacco | 33 |
| 8.6.2.3. | Activity | 33 |
| 9. | STUDY PROCEDURES | 34 |
| 9.1. | Screening and Baseline Assessments | 39 |
| 9.1.1. | Informed Consent | 39 |
| 9.1.2. | Demographics | 39 |
| 9.1.3. | Medical History | 39 |
| 9.1.4. | Eligibility Review | 40 |
| 9.1.5. | Drug and Alcohol Screening | 40 |
| 9.1.6. | Serology Testing | 40 |
| 9.1.7. | Prior and Concomitant Medication | |
| 9.1.8. | Other Screening Assessments | 40 |
| 10. | PHARMACOKINETICS | 41 |
| 10.1. | Pharmacokinetic Sampling | 41 |
| 10.1.1. | Blood Samples | 41 |
| 10.1.2. | Pharmacokinetic Evaluation | 41 |
| 10.2. | Pharmacokinetic Analytical Methodology | 41 |
| 11. | PHARMACODYNAMICS | 42 |
| 11.1. | Pharmacodynamic Sampling | 42 |
| 11.1.1. | Blood Samples | |
| 11.1.2. | Pharmacodynamic Evaluation | |
| 11.1.3. | Pharmacodynamic Analytical Methodology | |
| 12 | SAFETY ASSESSMENTS | 44 |

| 12.1. | Vital Signs | 44 |
|-----------|-------------------------------------------------------|----|
| 12.2. | Physical Examination | 44 |
| 12.3. | Electrocardiograms | 44 |
| 12.4. | Laboratory Assessments | 45 |
| 12.5. | Injection Site Assessment | 45 |
| 12.6. | Adverse Events | 46 |
| 12.6.1. | Definitions | 46 |
| 12.6.1.1. | Adverse Event | 46 |
| 12.6.1.2. | Adverse Reaction | 46 |
| 12.6.1.3. | Serious Adverse Event | 46 |
| 12.6.1.4. | Pre-treatment Adverse Event | 47 |
| 12.6.1.5. | Treatment-Emergent Adverse Event | 47 |
| 12.6.1.6. | Unexpected Adverse Reaction | 47 |
| 12.6.2. | Adverse Event Collection, Assessment and Reporting | 47 |
| 12.6.2.1. | Observation Period for Assessment of Adverse Events | 47 |
| 12.6.2.2. | Parameters for Adverse Events Collection | 47 |
| 12.6.3. | Assessment of Event Severity | 48 |
| 12.6.4. | Relationship to Study Treatment | 49 |
| 12.6.5. | Serious Adverse Event Reporting | 49 |
| 12.7. | Drug-Induced Liver Injury Monitoring | 50 |
| 12.7.1. | Pregnancy | 50 |
| 12.7.2. | Accidental Overdose, Medication Error, or Drug Misuse | 51 |
| 13. | OTHER ASSESSMENTS | 52 |
| 13.1. | Euglycemic Clamp Procedure | 52 |
| 14. | STATISTICAL ANALYSIS | 53 |
| 14.1. | Determination of Sample Size | 53 |
| 14.2. | Analysis Populations | 53 |
| 14.3. | Pharmacokinetic Analysis | 54 |
| 14.4. | Pharmacodynamic Analysis | 55 |
| 14.5. | Safety Analysis | 55 |
| 14.6. | Other Analyses | 56 |
| 14.7. | Interim Analysis | 56 |
| 14.8. | Data Monitoring Committee | 56 |

| 15. | STUDY MANAGEMENT | 57 |
|---|---|---|
| 15.1. | Approval and Consent | 57 |
| 15.1.1. | Compliance with Laws and Regulations | 57 |
| 15.1.2. | Institutional Review Board/Independent Ethics Committee | 57 |
| 15.1.3. | Informed Consent Process | 57 |
| 15.1.3.1. | Consent and Other Informational Documents Provided to Participants | 57 |
| 15.1.3.2. | Consent Procedures and Documentation | 57 |
| 15.2. | Study Discontinuation and Closure | 58 |
| 15.3. | Confidentiality and Privacy | 58 |
| 15.4. | Future Use of Stored Specimens and Data | 59 |
| 15.5. | Safety Oversight | 59 |
| 15.6. | Clinical Monitoring | 59 |
| 15.7. | Quality Assurance and Quality Control | 59 |
| 15.8. | Data Handling and Record Keeping | 60 |
| 15.8.1. | Data Collection and Management Responsibilities | 60 |
| 15.8.2. | Study Records Retention | 60 |
| 15.9. | Protocol Amendment and Protocol Deviation | 60 |
| 15.9.1. | Protocol Amendment | 60 |
| 15.9.2. | Protocol Deviations | 61 |
| 15.10. | Ethical Considerations | 61 |
| 15.11. | Financing and Insurance | 61 |
| 15.12. | Publication Policy | 61 |
| 15.13. | Conflict of Interest Policy | 62 |
| 16. | REFERENCES | 63 |
| 17. | APPENDICES | 64 |
| APPENDI | IX 1. CONTRACEPTION DEFINITIONS AND REQUIREMENTS | 65 |
| APPENIDI | IX 2 PROTOCOL AMENDMENTS | 67 |

# LIST OF TABLES

| Table 1. | Objectives and Endpoints | 19 |
|---|---|---|
| Table 2 | Study Treatments | |
| Table 3. | Schedule of Assessments | |
| Table 4. | Pharmacokinetic, Pharmacodynamic, C-Peptide, and Glucose Sampling Schedule | 38 |
| Table 5 | Pharmacokinetic Parameters | 41 |
| Table 6 | Pharmacodynamic Parameters | 42 |
| Table 7 | Laboratory Assessments | 45 |
| Table 8 | Classification of Adverse Events by Relationship to Study Treatment | 49 |
| Table 9. | Studies Referenced for Sample Size Assumptions | 53 |
| | LIST OF FIGURES | |
| Figure 1. | Study Design | 22 |
| Figure 2 | Investigational Product Description | 27 |
| Figure 3 | Control Treatment | 28 |

## 3. LIST OF ABBREVIATIONS

| Abbreviation | Expanded Term |
|--------------|------------------------------------------------|
| AE | adverse event |
| ADL | activities of daily living |
| ALT | alanine aminotransferase |
| Anti-HBc | antibody to hepatitis B core antigen |
| AST | aspartate aminotransferase |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CL/F | clearance |
| CMP | Clinical Monitoring Plan |
| COVID-19 | Coronavirus disease 2019 |
| CRO | Contract Research Organization |
| CRU | clinical research unit |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTR | Clinical Trial Regulation |
| CV | coefficient of variance |
| ECG | electrocardiogram |
| eCRF | Electronic Case Report Form |
| EOS | end of study |
| EU | European Union |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GIR | glucose infusion rate |
| HBsAg | hepatitis B surface antigen |
| HCV | hepatitis C virus |
| HIV | human immunodeficiency virus |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| ID | identification |
| IgM | immunoglobulin M |
| INR | international normal ratio |
| IRB | Institutional Review Board |
| MRT | mean residence time |
| NCI | National Cancer Institute |
| PD | pharmacodynamic |
| PI | Principal Investigator |
| PK | pharmacokinetic |
| QC | Quality Control |
| QTcF | QT-interval corrected by Fridericia's formula |

| SAE | serious adverse event |
|------|---------------------------------------------|
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous(ly) |
| SD | standard deviation |
| SmPC | Summary of Product Characteristics |
| SOP | Standard Operating Procedure |
| t½.z | apparent terminal elimination half-life |
| TEAE | treatment-emergent adverse events |
| ULN | upper limit of normal |
| US | United States |
| USPI | United States Prescribing Information |
| V/F | volume of distribution |
| λz | apparent terminal elimination rate constant |

Note: Definitions of pharmacokinetic (PK) and pharmacodynamic (PD) parameters are provided in Section 10.1.2 and Section 11.1.2.

#### 4. INTRODUCTION

Insulin therapy is essential for the treatment of diabetes mellitus Type 1 and is sometimes used in diabetes mellitus Type 2. Insulin aspart is a short-acting insulin. The onset of action is approximately fifteen minutes, the peak action is reached in 45–90 minutes, and the duration is 3–5 hours.

Currently available mealtime insulin analogues, while associated with a lower risk of hypoglycemia, are expensive (Ampudia Blasco, 2020). Insulin aspart is a rapid-acting insulin marketed as NovoLog® in the United States (US) and NovoRapid® in the European Union (EU). It has a faster onset and a shorter duration of action, resulting in postprandial glycemic control by means of lowering the total glucose excursion following a meal.

Biosimilar insulins should offer the advantages of insulin analogues at reduced costs.

## 4.1. Background on NKF-INS(A)

As a proposed biosimilar to insulin aspart, NKF-INS(A) has the potential to address the critical unmet need for cost-effective insulins, in patients with diabetes.

To demonstrate biosimilarity compared to US-approved and EU-authorized insulin aspart, a comparative clinical pharmacology study between the proposed insulin aspart test product (NKF-INS(A)) and both US-NovoLog® and EU-NovoRapid® reference products is required. This study should provide a time-concentration profile and a time-action profile over the duration of action of each product based on reliable measures of systemic exposure and glucose response.

As a proposed biosimilar to insulin aspart, NKF-INS(A) has the same amino acid sequence as NovoLog® and NovoRapid®. Insulin aspart is homologues with regular human insulin with the exception of a single substitution of the amino acid proline by aspartic acid in position B28. NKF-INS(A) is produced by recombinant DNA technology utilizing *Escherichia coli* whereas NovoLog® and NovoRapid® are produced in *Saccharomyces cerevisiae* by recombinant DNA technology. NKF-INS(A) has the empirical formula of C<sub>256</sub>H<sub>381</sub>N<sub>65</sub>O<sub>79</sub>S<sub>6</sub> and has a molecular weight of 5822.6 Da.

As in human insulin, insulin aspart contains two interchain disulfide bonds, and one intrachain disulfide bond.

The primary activity of insulin aspart is the regulation of glucose metabolism. Insulins, including insulin aspart, bind to the insulin receptors on muscle and fat cells and lower blood glucose by facilitating the cellular uptake of glucose and simultaneously inhibiting the output of glucose from the liver.

This is the first clinical study of NKF-INS(A) drug product.

## 4.1.1. Preliminary Analytical Similarity Study for Program Feasibility

To confirm the feasibility with the Food and Drug Administration (FDA) for the licensure in the US of insulin aspart as a biosimilar to US-licensed US-NovoLog® through the 351(k) pathway, a preliminary analytical similarity study was conducted between the reference product and US-insulin aspart early development drug substance lots, utilizing a subset of quality attributes to be included in the full analytical similarity test panel. Three lots of US-licensed NovoLog® were

included and three insulin aspart early development drug substance lots were included in this similarity study. The most critical quality attributes that were not likely to be significantly impacted by the drug product fill/finish process and container closure were included in this study.

The preliminary analytical similarity study results demonstrated that insulin aspart is highly similar to the US-reference product in both physicochemical and biological characteristics, therefore further development of insulin aspart as a biosimilar to US-NovoLog<sup>®</sup> is feasible.

No other nonclinical animal studies or clinical studies have been completed for insulin aspart.

## 4.2. Clinical Benefits/Risks of NKF-INS(A)

The safety profile of NKF-INS(A) has not been evaluated in humans. Based on currently approved insulin aspart products, side effects include allergic reactions, hypoglycemia, hypokalemia, and weight gain. Recognizing that NKF-INS(A) is a biosimilar product, no additional risks are expected; however, participants will be closely monitored throughout the study for side effects.

Details regarding known or anticipated benefits and risks, as well as reasonably anticipated adverse events (AEs) for NKF-INS(A) are provided in the Investigator's Brochure.

## 4.3. Study Rationale

Despite advances in diabetes mellitus care, there remains a critical unmet need for cost-effective insulins in many markets.

As a biosimilar to insulin aspart, NKF-INS(A) has the potential to address this unmet medical need in patients with diabetes mellitus. In order to demonstrate biosimilarity of NKF-INS(A) to EU-NovoRapid® and US-NovoLog®, a Phase 1 study will evaluate the PK and PD of NKF-INS(A) to the reference products using a euglycemic clamp technique in healthy male volunteers.

#### 4.4. Dose Rationale

NKF-INS(A), EU-NovoRapid<sup>®</sup> and US-NovoLog<sup>®</sup> will be administered as a 0.3 U/kg single subcutaneous (SC) dose in the periumbilical area. US-NovoLog<sup>®</sup> and EU-NovoRapid<sup>®</sup> are dosed between 0.5 U/kg/day and 1.0 U/k/day to patients with diabetes mellitus (Novolog US Prescribing Information [PI], 2008). Given this study will recruit healthy male participants, a dose of 0.3 U/kg was selected and aligned with similar trials of aspart analogues (Chen et al, 2023; Drai et al, 2022; Hövelmann et al, 2021).

NKF-INS(A) dosage is individualized based on the route of administration, and the participant's metabolic needs, blood glucose monitoring results, and glycemic control goal. For the purposes of the clinical study, the participant will receive a single dose of 0.3 U/kg SC by injection in the periumbilical area in three treatment sequences.

## 5. STUDY OBJECTIVES AND ENDPOINTS

Objectives and related endpoints are described in Table 1.

Table 1. Objectives and Endpoints

| Objectives | |
|---|---|
| Primary | |
| To compare the PK of NKF-INS(A) to US-approved and EU-authorized insulin aspart to demonstrate PK similarity for insulin aspart. | <ul> <li>Aspart concentration-time curve from 0 to 12 hours (AUC<sub>0-t</sub>)</li> <li>Maximum observed insulin aspart concentration (C<sub>max</sub>)</li> </ul> |
| To compare the PD of NKF-INS(A) to<br>US-approved and EU-authorized insulin<br>aspart injection by examining GIR profiles<br>after a single SC dose. | <ul> <li>Area under the GIR-time curve from 0 to 12 hours (AUCGIR<sub>0-t</sub>)</li> <li>Maximum GIR (GIR<sub>max</sub>) of glucose</li> </ul> |
| Secondary | |
| To evaluate additional PK parameters of<br>NKF-INS(A) compared to US-approved and<br>EU-authorized insulin aspart. | • PK parameters for serum insulin aspart concentrations: AUC <sub>0-4h</sub> , AUC <sub>0-6h</sub> , AUC <sub>6-12h</sub> , AUC <sub>0-12h</sub> , T <sub>max</sub> , AUC <sub>0-∞</sub> |
| | Time to half-maximum before C <sub>max</sub> (t50%-early) |
| | • Time to half-maximum after C <sub>max</sub> (t50%-late) |
| | • The terminal elimination half-life (t <sub>1/2</sub> ) |
| To evaluate additional PD parameters of<br>NKF-INS(A) compared to US-approved and<br>EU-authorized insulin aspart. | • AUCGIR from 0 to 4 hours (AUCGIR <sub>0-4h</sub> ), from 0 to 6 hours (AUCGIR <sub>0-6h</sub> ), and from 6 hours until the end of clamp (AUCGIR <sub>6-last</sub> ) |
| | Time to maximum glucose infusion rate (T <sub>max</sub> .GIR) |
| | Time to half-maximum glucose infusion rate<br>before GIR <sub>max</sub> (tGIR,50%-early) |
| | Time to half-maximum glucose infusion rate<br>after GIR <sub>max</sub> (tGIR,50%-late, indicator of end<br>of duration of action) |
| | <ul> <li>Time from study drug administration until the blood glucose concentration has decreased by at least 5 mg/dL from baseline (onset of action)</li> <li>The difference between tGIR,50%-late and the onset of action (duration of action)</li> </ul> |

| Objectives | |
|---|---|
| To assess the safety of NKF-INS(A). | AE assessments, (including injection site reactions), clinical laboratory investigations (hematology, clinical chemistry [including glucose], coagulation, and urinalysis), vital signs, physical examinations, 12-lead ECG, prior and concomitant medication assessments |
| Exploratory | |
| To assess endogenous insulin suppression<br>via C-peptide measurements, which includes<br>both corrected and uncorrected C-peptide<br>concentrations. | <ul> <li>Corrected and uncorrected C-peptide concentrations</li> <li>If possible, i.e., if the terminal phase of serum concentration-time profile has sufficient data points, apparent terminal elimination half-life (t½.z), apparent terminal elimination rate constant (λz), mean residence time (MRT), clearance (CL/F), and volume of distribution (V/F) will be calculated</li> </ul> |

Abbreviations: AE = adverse events; ECG = electrocardiogram; EU = European Union; GIR = glucose infusion rate; PD = pharmacodynamic; PK = pharmacokinetics; SC = subcutaneous; US = United States

#### 6. INVESTIGATIONAL PLAN

## 6.1. Description of Overall Study Design and Plan

The NKF-INS(A) clinical program is designed to demonstrate biosimilarity to the US and EU-insulin aspart (EU-NovoRapid<sup>®</sup>, and US-NovoLog<sup>®</sup>) by comparing the PK and PD of NKF-INS(A) to the reference products after a single SC dose.

Study NKF-INS(A)-101 is a Phase 1, 12-hour euglycemic glucose clamp study conducted using a randomized, double-blind, three-period, three-treatment, six-sequence, crossover design. The study will compare single doses of the proposed insulin biosimilar (NKF-INS(A)) with respective EU- and US-reference products in healthy male participants.

Written informed consent will be obtained from all participants, and the study will be conducted in accordance with the principles of Good Clinical Practice (GCP) as defined by the International Conference of Harmonization (ICH).

The study will consist of:

- a screening period of up to 4 weeks (Days -28 to -1),
- three treatment periods each consisting of 1-day dose administrations and euglycemic clamp periods (periods 1, 2, and 3) separated by a washout period of 3-14 calendar days between treatment periods 1 and 2, and a washout period of 5-21 calendar days between treatment periods 2 and 3, and
- a follow-up period of 2-11 days after last dose.

The entire study duration will be a maximum of 11 weeks.

Three insulin products (NKF-INS(A), EU-NovoRapid®, and US-NovoLog®) will be administered over three treatment periods. Upon admission to the clinical research unit (CRU) on Day -1, participants will be randomized to one of six treatment sequences in a 1:1:1:1:1 ratio, receiving a single SC dose of 0.3 U/kg administration of one of the three study drugs on each dosing day.

A 12-hour euglycemic glucose clamp will be conducted using a manual clamp technique, which will monitor the subject's blood glucose and administer glucose infusion rate (GIR) to maintain blood glucose close to the target blood glucose concentration. The clamp procedure will be initiated, maintained, and terminated, in accordance with the site standard operating procedures (SOPs). The participant's blood glucose will be maintained within a pre-defined target window per site SOP and clinical judgment for the participant by manually adjusting the GIR.

Blood samples will be collected at pre-specified intervals before and up to 12 hours after dosing for measurement of blood glucose, serum insulin, and C-peptide.

Fifty-four healthy male participants are planned to be enrolled in the study to have at least 36 evaluable participants.

The following steps will be taken to minimize variability:

- Prior to each dosing, participants will have been fasting for 10-12 hours
- Individual participants will be dosed at about the same time of day within each treatment period
- The injection site and technique will be standardized between treatment periods
- Any occurrence of a drop in glucose below 3.3 mmol/L will be recorded as this may induce counter-regulatory hormones

The study design schema is provided in Figure 1.

Figure 1. Study Design



Abbreviations: EU = European Union; US = United States

## **6.2.** Discussion of Study Design

Congruent to Draft Guidance "Clinical Immunogenicity Considerations for Biosimilar and Interchangeable Insulin Products", the Sponsor believes the aforementioned comparative analytical assessment demonstrates NKF-INS(A) is highly similar to EU-NovoRapid®, and US-NovoLog® and there is no residual uncertainty regarding immunogenicity. Therefore, in addition to the comparative analytical assessments, the Sponsor plans to conduct one Phase 1 study to demonstrate PK similarity to reference products to provide a totality of evidence for biosimilarity for licensure.

The design of the study was chosen as both FDA and European Medicines Agency recognize the clamp technique as the most reliable method for qualifying the PK and PD proprieties of a novel biosimilar. Clamp technique is used to rapidly attain the required blood glucose levels and maintain it at target levels (Heinemann et al, 2023).

## 6.3. End of Study

A participant will have fulfilled the requirements for study completion if/when the participant has completed all three treatment periods and the end of study (EOS) visit within 2-11 days after last administration of the study drug.

The EOS is defined as the date of the last visit for the last participant in the study/last scheduled procedure shown in the schedule of assessments (Table 3).

## 6.4. Criteria for Early Study Termination

The Sponsor reserves the right to close a study site or terminate the study at any time for any reason. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study site closure visit has been performed.

The Investigator may initiate study site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the Sponsor or Investigator may include but are not limited to:

- Failure of the Investigator to comply with the protocol, requirements of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) or local health authorities, the Sponsor's procedures, or ICH GCP guidelines, or contractual agreement.
- Inadequate recruitment of participants by the Investigator.
- Discontinuation of further development of NKF-INS(A).

The IRB/IEC and regulatory authorities will be informed about the reason and time of the termination according to applicable laws and regulations. If the study is terminated prematurely, Investigators will inform their participants.

#### 7. SELECTION OF STUDY POPULATION

#### 7.1. Inclusion Criteria

Individuals must meet all of the following inclusion criteria to be included in the study:

- 1. Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the participant.
- 2. Healthy male participants.
- 3. Age between 18 and 50 years, both inclusive.
- 4. Body Mass Index between 18.5 and 29.0 kg/m<sup>2</sup>, both inclusive.
- 5. Body weight  $\geq$  50 kg.
- 6. Fasting plasma glucose concentration  $\leq 5.5$  mmol/L at screening.
- 7. Considered generally healthy upon completion of medical history, physical examination, vital signs, ECG, and analysis of laboratory safety variables, as judged by the Investigator.
- 8. Willing and able to comply with scheduled visits, treatment plan, clinical laboratory tests, and other study procedures including lifestyle considerations.
- 9. Participants must agree to use condoms during sexual intercourse. Additionally, female partners of male participants should use highly effective contraception. All contraceptive measures apply from screening until 90 days after study treatment. Male participants must refrain from donating or banking sperm for 90 days after administration of study treatment.
- 10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.

#### 7.2. Exclusion Criteria

Individuals will be excluded from participation if they meet any of the following criteria:

- 1. Positive for human insulin antibodies at Screening.
- 2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.
- 3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.
- 4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.

- 5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.
- 6. Have clinically relevant history of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.
- 7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.
- 8. Clinically significant abnormal ECG at screening.
- 9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load.
- 10. Show evidence of significant active neuropsychiatric disease.
- 11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year.
- 12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment.
- 13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening.
- 14. Have positive test results for hepatitis B surface antigen (HBsAg), immunoglobulin M (IgM) antibody to hepatitis B core antigen (anti-HBc), or hepatitis C virus (HCV) antibodies at screening.
- 15. Intend to use over-the-counter medication within 7 days or prescription medication within 14 days prior to dosing (apart from vitamin/mineral supplements, occasional paracetamol, thyroid replacement).
- 16. Have donated blood or had a blood loss of 450 mL 3 months prior to study enrollment.
- 17. Have an average weekly alcohol intake that exceeds 21 units per week or is unwilling to stop alcohol consumption from 48 hours prior to each dosing until being discharged from the CRU.

## 7.3. Rescreening

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently entered into the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse event (SAE).

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened only once, at the discretion of the Investigator.

The participant must be reconsented and a new screening number will be assigned. Also, a new informed consent form (ICF) must be signed if updates have been made since signing of the first ICF.

## 7.4. Study Withdrawal, Removal, and Replacement of Participants

Participants may withdraw from the study at any time with or without reason. The Investigator also has the right to discontinue or terminate participants from the study in the event of concomitant disease, AEs, or any reason that would benefit the participant (see Section 8.4).

If a participant withdraws from the study for any reason, the study site must immediately notify the clinical monitor. The date and the reason for study discontinuation must be recorded in the electronic case report form (eCRF). Participants who discontinue early, irrespective of the reason for discontinuation from the study, will be asked to complete the EOS assessments at the time of the participant's withdrawal, as outlined in the schedule of assessments (Table 3).

If a participant withdraws from the study, he may request destruction of any samples taken and not tested, and the Investigator must document this in the site study records.

Additionally (as described in Section 6.4), the Sponsor may stop the study at any time for safety, regulatory, legal, or other reasons aligned with GCP. This study may be terminated at the discretion of the Sponsor or any regulatory agency. An Investigator may elect to discontinue or stop the study at his or her study site for any reason, including safety or low enrollment.

## 7.4.1. Replacement of Participants

Participants who sign the ICF and are randomized but not treated may be replaced at the discretion of the Sponsor.

#### 8. TREATMENTS

A list of study treatments used in this study is provided in Table 2.

**Table 2** Study Treatments

| Agent | Use |
|---|---|
| NKF-INS(A) | Investigational agent |
| US-NovoLog®, and | Indicated to improve glycemic control in adults and children with diabetes |
| EU-NovoRapid® Flex | mellitus |
| Pen | |

Source: NovoLog® United States Prescribing Information (USPI); NovoRapid Summary of Product Characteristics

## 8.1. Study Treatment Description

NKF-INS(A), US-NovoLog® and EU-NovoRapid® is intended to be administered as a 0.3 U/kg single dose SC in the periumbilical area.

US-NovoLog® and EU-NovoRapid® will be supplied by Novo Nordisk, Plainsboro, NJ, US.

NKF-INS(A) is a clear and colorless solution.

NKF-INS(A) is supplied in a disposable pen (with cartridge) containing 300 U/3mL; 1 mL solution contains 100 units of NKF-INS(A), equivalent to 3.5 mg. The disposable pen syringe device is a BD Vystra Disposable Pen sourced commercially (Figure 2).

Figure 2 Investigational Product Description

BD Vystra™ Disposable Pen



Note: Colors shown are approximate. Appearance may differ based on individual computer monitor or printer settings.

US-NovoLog® and EU-NovoRapid® is supplied in a disposable pen syringe containing 300 U/3mL (NovoLogâ United States Prescribing Information (USPI); NovoRapid Summary of Product Characteristics[SmPC]); 1 mL solution contains 100 units of insulin aspart equivalent to 3.5 mg. The disposable pen is a proprietary device with a NovoFine needle (Figure 3).

#### Figure 3 Control Treatment



Diagram A FlexPen Prefilled Syringe

#### NovoFine® needle



Diagram B NovoFine needle

#### 8.1.1. Preparation, Handling, and Disposal

The preparation of NKF-INS(A), US-NovoLog® and EU-NovoRapid® will be conducted in accordance with the Pharmacy Manual.

Procedures for proper handling and disposal should be followed in compliance with the SOPs of the site.

#### 8.1.2. Product Labeling and Packaging

NKF-INS(A), US-NovoLog® and EU-NovoRapid® will be labeled to meet country-specific regulatory requirements.

Refer to the Pharmacy Manual for packaging and labeling information.

#### 8.1.3. Administration

NKF-INS(A), US-NovoLog® and EU-NovoRapid® will be administered as a single dose via the SC route (refer to Section 8.2). Device-related events or complaints should be reported to the Sponsor in accordance with the Pharmacy Manual.

#### **8.1.4. Storage**

Refer to the Pharmacy Manual for information regarding storage, handling, and administration of NKF-INS(A), US-NovoLog<sup>®</sup> and EU-NovoRapid<sup>®</sup>.

Before opening (unpunctured), NKF-INS(A) should be stored at 2 °C to 8 °C (36 °F to 46 °F) and protected from heat and light until the time of use. The drug product must not be frozen or placed adjacent to the refrigerator cooling element.

During use (punctured), NKF-INS(A) should be stored below 30 °C (86 °F) for up to 28 days and should not be exposed to excessive heat or sunlight. Do not freeze and do not draw into a syringe for later use. Pen cap should be kept on the pen in order to protect from light.

Always remove and discard the needle after each injection of NKF-INS(A) pen. Pens are considered single use.

The shelf life during use for US-NovoLog® and EU-NovoRapid® is 28 days when stored below 30 °C (86 °F). The unpunctured disposable pen can be used until their expiry date if stored at 2 °C to 8 °C (36 °F to 46 °F). NKF-INS(A) is being studied on an ongoing stability program and is tested at regular intervals to establish shelf life.

## 8.2. Dosage Schedule

Upon admission to the CRU on Day -1, participants will be randomized on Day 1 to one of six treatment sequences in a 1:1:1:1:1 ratio, receiving a single SC dose of 0.3 U/kg administration of one of the three study drugs on each dosing day.

The insulin products will be administered using an euglycemic glucose clamp at a targeted blood glucose concentration. The euglycemic glucose clamp will be conducted using a clamp technique. The glucose clamp device will manually adjust the infused GIR to maintain the target blood glucose concentration based on the actual measured blood glucose concentration and the degree of variability in the previous minute.

Blood samples will be collected at pre-specified intervals before and up to 12 hours after dosing for measurement of blood glucose, serum insulin, and C-peptide.

Participants will visit the study site for 3 single-dose periods with specified washouts (3-14 days between treatment periods 1 and 2; and 5-21 days between treatment periods 2 and 3). The entire duration of the study will be a maximum of 11 weeks.

# 8.3. Measures to Minimize Bias: Study Treatment Assignment and Blinding

#### 8.3.1. Method of Study Treatment Assignment

Participants will be assigned a screening identification (ID) number when providing informed consent. A participant ID will be provided on Day -1. A participant ID consists of a site ID and a participant number that uniquely identifies each participant.

On Day 1, participants will be randomly allocated to study treatment sequence according to a pre-specified randomization scheme prepared by an independent statistician (refer to Section 8.2).

#### 8.3.2. Blinding

All participants, Investigators, and study personnel involved in the conduct of the study will be blinded to treatment assignment with the exception of unblinded statistician, programmer, pharmacists, and drug administrator.

Because study drug and comparator differ slightly in appearance, the study drug will be prepared by an unblinded pharmacist and administered by an unblinded administrator, while the participant is blindfolded. The used pen will be returned to the packaging and reconciliation will be completed by the unblinded pharmacist.

The unblinded study personnel will not participate in study procedures or data analysis prior to unblinding of the study data.

The following controls will be employed to maintain the double-blind status of the study:

The randomization list will be kept within the Clinical Data Management System and role-based access will prevent any unauthorized personnel from accessing the blinded information. The pharmacist will have access to the randomization list for dispensing purposes.

- To manage the participant's condition in case of a medical emergency, the Investigator will be able to break the blind for a specific participant, using the Clinical Data Management System, to know whether a participant received NKF-INS(A), US-NovoLog® and EU-NovoRapid®. In order to break the blind, the Investigator will have to provide a reason for doing so. All relevant data including the responsible individual, the date, the time, and the reason for breaking the blind will be captured electronically within audit trail of the Clinical Data Management System. The Sponsor will be informed in case of unblinding.
- Extra measures (where relevant) will be put in place to maintain the blind during dosing, e.g., blindfolding of participants, presenting the study treatments as identical in appearance where possible, double-blind labelling, unblinded personnel to administer study treatment.

#### 8.4. Treatment Modifications and Discontinuations

Dose reductions and adjustments are not permitted; any dose reductions and adjustments that occur will be recorded and considered protocol deviations.

Delays and omissions of study treatment administration because of medical or nonmedical reasons are not permitted. All delays and omissions of study treatment that occur during the study will be recorded and considered protocol deviations.

A participant may be discontinued from the study at any time for reasons including, but not limited to, the following:

- AE and/or SAEs in the judgment of the Investigator that may prevent the participant from continuing participation in the study.
- Participant withdrawal of consent (at any time, a participant's participation in the study may be terminated at their request).
- On the basis of the Investigator's clinical judgment.
- General or specific changes in the participant's condition that render them ineligible for further treatment according to the inclusion/exclusion criteria.
- Participant fails to adhere to the protocol requirements (e.g., study treatment noncompliance).
- Lost to follow up: the participant stopped coming for visits and study personnel were unable to contact the participant.

Note: In cases in which the participant is deemed lost to follow up, prior to this designation, the Investigator (or designee) must make every effort to make contact with the participant (e.g., telephone calls, certified letter to the participant's last known mailing address, or local equivalent methods, and efforts to reach the participant's emergency contact). The site will make 3 attempts to regain contact with the participant. These contact attempts must be documented in the participant's medical records.

Any participant who discontinues from the study will be asked to return to the clinic for an EOS visit that includes the assessments as shown in the schedule of assessments (Table 3). The reason and date for the participant's discontinuation from the study must be recorded in the eCRF.

## 8.5. Treatment Accountability and Compliance

The pharmacist or other designated individual will maintain records of study drug delivered to the study site, the inventory at the study site, the distribution to and use by each participant, and the return of materials to the Sponsor for storage or disposal/destruction of materials at the study site. These records must include dates, quantities, lot/batch/serial numbers, expiration dates, storage temperature log, and unique code numbers assigned to the study drug and study participants.

Investigators/designee will maintain records that adequately document that the participants were provided with the correct study treatment and reconcile the products received from the drug dispensing center. Investigational product will not be returned to the Sponsor or disposed of until accountability has been fully monitored.

Administration of the study treatment will be supervised by unblinded study site personnel to ensure compliance. An unblinded monitor will periodically review the study records to ensure compliance. Discontinuation for noncompliance is at the Investigator's discretion and is to be noted in the eCRF.

Cases of accidental overdose or medication error, along with any associated AEs, should be reported as described in Section 12.6.2.

# 8.6. Prior and Concomitant Therapy and Other Restrictions During the Study

#### **8.6.1.** Prior and Concomitant Medications

Medications taken by or administered to the participant for the period before screening will be recorded in the eCRF as prior medications. Restricted prior therapies include over-the-counter medication within 7 days or prescription medication within 14 days prior to dosing (apart from vitamin/mineral supplements, occasional paracetamol, thyroid replacement, or birth control methods).

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) other than NKF-INS(A), US-NovoLog® and EU-NovoRapid® that the participant is receiving at the time of enrollment, or receives during the study, must be recorded in the eCRF as concomitant medications along with:

• Reason for use

- Dates of administration including start and end dates
- Dosage information including dose, regimen, route, and frequency

The participant must be told to notify the investigational site about any new medications taken after administration of the study treatment.

All previous and on study Coronavirus disease 2019 (COVID-19) vaccinations should be recorded in the eCRF.

The Medical Monitor should be contacted if there are any questions regarding prior or concomitant therapy.

#### **8.6.1.1.** Permitted Concomitant Medications and Therapies

Other than those medications explicitly prohibited (Section 8.6.1), concomitant medication decisions will be left to the discretion of the Investigator.

### **8.6.1.2.** Prohibited Concomitant Medications and Therapies

Participants must be instructed not to take any medications, including over-the-counter products, without first consulting with the Investigator.

If the participant has received any other investigational drug within 3 months before the administration of study treatment, he will not be eligible for this study.

No prophylactic medication, treatments, or procedures will be administered during the study period, unless at the discretion of the Investigator.

### 8.6.1.3. Advisory on COVID-19 Vaccination and Risk Assessment

The COVID-19 pandemic is an ongoing pandemic with varying impact at any time in different geographies worldwide (World). It is recommended that participants and their investigators discuss on an individual basis the benefits and risks of COVID-19 vaccination in the context of their prior vaccination history and consider the vaccinations approved by national regulatory agencies, as well as COVID-19 vaccination guidance from scientific and medical associations.

The following recommendations should be considered for the study:

- Participants with prior COVID-19 vaccination may be allowed to enter the study with a washout period of at least 7 days since the last COVID-19 vaccine dose.
- Administration of a COVID-19 vaccine during participation in the study should be documented as a concomitant medication (Section 8.6.1).
- Previous administration(s) of COVID-19 vaccine should be documented in the prior and concomitant medication form.

#### 8.6.2. Other Restrictions During the Study

## 8.6.2.1. Meals and Dietary Restrictions

For all treatment periods, participants will fast for 10-12 hours prior to dosing and until the glucose clamp procedure is completed, after which participants will receive a meal. There is no restriction on water during the fasting periods of the study. When not in CRU subjects will be encouraged to follow their normal diets. Grapefruit juice is an inhibitor of the CYP3A4 enzyme but CYP3A4 does not play a role in the metabolism of insulin aspart thus it is not mentioned.

#### 8.6.2.2. Caffeine, Alcohol and Tobacco

No alcohol will be allowed 48 hours before each dose and for the duration of each CRU visit.

Participants should refrain from caffeine-containing food/beverages for at least 24 hours before each dose and through the duration of visit.

Smoking of tobacco products, nicotine replacements etc., will not be permitted during the confinement period.

#### **8.6.2.3.** Activity

Participants are encouraged to maintain their regular exercise habits; however, they should not undertake vigorous or prolonged exercise within 48 hours prior to dosing. Strenuous exercise is not allowed throughout the entire study.

#### 9. STUDY PROCEDURES

Assessments and their timing to be performed are outlined in the schedule of assessments (Table 3).

See Sections 10, 11, 12, and 13 for additional details regarding PK, PD, safety, and other assessments, respectively.

The Investigator may, at his or her discretion, arrange for a participant to have an unscheduled assessment, especially in the case of AEs that require follow up or are considered by the Investigator to be possibly related to the use of study treatment. The unscheduled visit page in the eCRF must be completed for all unscheduled assessments.

 Table 3.
 Schedule of Assessments

| | Screening | Screening Euglycemic Clamp Procedure Treatment Periods 1-3 <sup>1</sup> | | | EOS Visit |
|---|---|---|---|---|---|
| Assessment | -28 to -1 Days Priorto<br>Treatment Period 1 | Day -1 | Clamp Procedure Starting the Morning of Day 1 for 12 Hours <sup>2</sup> | Post-<br>Clamp<br>(Day 2) | Within 2-11 Days After Last Administration of Study Drug |
| Informed consent | X | | | | |
| Demographic data <sup>3</sup> | X | | | | |
| Alcohol and tobacco consumption patterns | X | | | | |
| Medical and medications<br>history <sup>4</sup> | X | X | | | |
| Inclusion/exclusion criteria | X | X | | | |
| Admission to CRU <sup>5</sup> | | X | | | |
| Randomization | | | $X^6$ | | |
| Discharge from CRU | | | | X | |
| Height/weight <sup>7</sup> | X | X | | | |
| Physical examination <sup>8</sup> | X | | | | X |
| Vital signs <sup>9</sup> | X | | X | X | X |
| 12-lead ECG | X | | | | X |
| Hematology <sup>10</sup> | X | | | | X |
| Clinical chemistry <sup>11</sup> | X | | | | X |
| Blood coagulation <sup>12</sup> | X | | | | |
| Serology tests<br>(HBsAg, IgM anti-HBc, HCV,<br>HIV) <sup>13</sup> | X | | | | |
| Urinalysis <sup>14</sup> | X | | | | |
| Urine screen for drugs of abuse 15 | X | X | | | |
| Alcohol breath test <sup>16</sup> | X | X | | | |
| Human insulin antibodies | X | | | | |
| Oral glucose tolerance test <sup>17</sup> | X | | | | |
| Study drug administration <sup>18</sup> | | | Day 1 at time = 0 hours/0 min | | |
| Injection site assessment <sup>19</sup> | | | X | | X |
| GIR | | | X | | |
| Adverse events | , | | | | <b>——</b> |
| | Screening | Euglycem | EOS Visit | | | |
|---|---|---|---|---|---|--|
| | | | | | Within 2-11 Days | |
| Assessment | | | Clamp Procedure | Post- | After Last | |
| | -28 to -1 Days Priorto | | Starting the Morning of Day 1 for | Clamp | Administration of | |
| | Treatment Period 1 | Day -1 | 12 Hours <sup>2</sup> | (Day 2) | Study Drug | |
| Concomitant medications | | | | | <b>→</b> | |
| PK, PD, C-peptide, and glucose sampling (see Table 4) | | | | | | |

Abbreviations: ALP = alkaline phosphatase; ALT = alanine aminotransferase; anti-HBc = antibody to hepatitis B core antigen; aPTT = activated partial thromboplastin time; AST = aspartate aminotransferase; CRU = clinical research unit; ECG = electrocardiogram; EOS = end of study; GGT = gamma-glutamyl transferase; GIR = glucose infusion rate; Hb = hemoglobin; HBsAg = hepatitis B surface antigen; HCT = hematocrit; HCV = hepatitis C virus; HIV = human immunodeficiency virus; IgM = immunoglobulin M; INR = international normalized ratio; MCH = mean corpuscular hemoglobin; MCV = mean corpuscular volume; PD = pharmacodynamic; PK = pharmacokinetic; PT = prothrombin time; RBC = red blood cell; WBC = white blood cell

- 1 There will be a washout period of 3-14 calendar days between treatment period 1 and 2, and a washout period of 5-21 calendar days between treatment periods 2 and 3.
- 2 The clamp procedure will be considered as ended if the 20% GIR is on zero (0) and the infusion pump has been stopped or the 12-hour mark is reached. Blood glucose concentration will be measured for 3 consecutive times for safety reasons, after the infusion pump is on zero (0).
- 3 Sex, race, year of birth, age, and ethnicity.
- 4 The recorded medical history will be updated, if necessary, at admission to treatment period 1.
- 5 Participants will be admitted to the CRU approximately 12 hours prior to dosing on Day -1.
- 6 Randomization will only be done on first sequence.
- 7 Body weight will be recorded at screening and on Day -1 of all treatment periods. The weight measured on Day -1 of treatment period 1 will be used for dosage calculations of insulin. Height will be recorded at screening only. 8 A full physical examination will include the following: Evaluation for jaundice, pallor (anemia), cyanosis, clubbing, edema and lymphadenopathy; skin evaluation; fundoscopy; ear, nose and throat; cardiovascular assessment; respiratory assessment; abdominal evaluation; musculoskeletal assessment; neurological assessment; other evaluations may be performed as deemed necessary by the Investigator. A full physical exam should be done at screening. A limited symptom-based physical exam may be done at timepoints thereafter.
- 9 Supine systolic and diastolic blood pressure, pulse, and respiratory rate will be recorded at screening, before administration of the study drug, at the end of the clamp (before discharge from the study center) and at the EOS visit. Body temperature (temporal or ear) will be recorded at screening and before administration of study drug (either standing or supine). All vital signs will be measured after the participant has been resting in a supine position for at least 5 minutes.
- 10 Hematology (ethylenediaminetetraacetic acid tubes): full and differential blood count, WBC count, RBC count, Hb, HCT, MCV, MCH, MCH concentration, absolute differential count (neutrophils, lymphocytes, monocytes, eosinophils and basophils), and platelets.
- 11 Clinical chemistry (serum separator tubes): potassium, sodium, urea, chloride, phosphorus, creatinine, calcium, albumin, total and direct bilirubin, creatine kinase, ALP, GGT, AST, ALT, lactate dehydrogenase, total cholesterol, triglycerides, and glucose.
- 12 Blood coagulation tests (citrated tubes): PT, aPTT, and INR.
- 13 Tests for HIV, HBsAg, IgM anti-HBc, and HCV, performed using commercially available test kits. Pre- and post-test counseling will be provided as appropriate.
- 14 Urinalysis (dipstick): appearance, bilirubin, glucose, ketone, specific gravity, blood, pH, protein, urobilinogen, nitrite, leucocytes. Abnormal urinalysis results may be repeated at the discretion of the Investigator.

- 15 A rapid, one-step screening test for simultaneous, qualitative detection of multiple drugs and drug metabolites will be used. Subjects with alleged false positive test results will be excluded from the study. However, a positive test may be repeated once at the discretion of the Investigator.
- 16 Alcohol breath test using a portable breath alcohol measuring device. The test will be performed at screening, at admission to each treatment period and at random. If any of these tests are positive, the subject will not be allowed further participation in the study.
- 17 Oral glucose tolerance test may be completed after all other eligibility has been determined. For participants who re-screen, oral glucose tolerance test does not need to be repeated if completed within the last 6 months.
- 18 From 1 hour before study drug administration until 3 hours post-dose, the injection site will be kept at a constant temperature. The time of injection is defined as time zero (0 hour/0 min) and marks the start of the clamp period, which will continue for up to 12 hours or until the GIR is 0 and blood glucose remains stable.
- 19 The injection site will be assessed at 1 min and 15 min post-dose on Day 1 and at the EOS visit. Reactions to the study drug injection will be documented using a numerical scoring system.

Table 4. Pharmacokinetic, Pharmacodynamic, C-Peptide, and Glucose Sampling Schedule

| | | re-dos<br>ninutes | | Post-dose (minutes) | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 20 | | _ | 1.0 | 20 | 20 | 40 | 5.0 | | | 00 | 105 | 120 | 125 | 1.50 | 100 | 210 | 240 | 200 | 600 | 720 |
| Sample | 60 | 30 | 0 | 5 | 10 | 20 | 30 | 40 | 50 | 60 | 75 | 90 | 105 | 120 | 135 | 150 | 180 | 210 | 240 | 300 | 600 | (12 hours) |
| Insulin (serum) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| C-peptide (serum) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood glucose | | | | Every 3 minutes | | | | | | ] | Every 5 | minute | s | | Ev | ery 10 1 | ninutes | | | | | |

# 9.1. Screening and Baseline Assessments

Standard study procedures will be performed at the timepoints indicated in the schedule of assessments (Table 3). A description of the study procedures is provided in the sections below.

#### 9.1.1. Informed Consent

Before performing any study-related procedures, the Investigator (or designee) will obtain written informed consent from the participant according to national legal regulations (see Section 15.1.3).

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened only once. Participants may be rescreened at the Investigator's discretion. The participant must be reconsented and a new screening number will be assigned. Also, a new ICF must be signed if updates have been made since signing of the first ICF.

To give the participant sufficient time to consider study participation, informed consent can be obtained before the screening visit. However, if the informed consent is obtained on the day of screening, then the time must be documented in the participant's chart to provide proof that consent was given before the first study-related screening procedure.

- The Investigator or their authorized representative will explain the nature of the study to the participant and answer all questions regarding the study.
- Participants will be informed that their participation is voluntary and will be required to sign a statement of informed consent that meets the requirements of the local regulations, the ICH guidelines, the IEC/IRB, or study site.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date (and time, if obtained on the day of screening) when the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must give new consent to each updated version of the ICF during their participation in the study.
- Each ICF must be personally dated and signed by the participant as well as by the Investigator (or designee).
- A copy of the ICF (or second original ICF per local regulations) must be provided to the participant. If the ICF is not taken by the participant, it will be archived with the participant's study documents.

#### 9.1.2. Demographics

Date of birth and/or age, sex at birth, race, ethnicity, and country will be recorded at screening in the eCRF.

### 9.1.3. Medical History

Medical history will be recorded at screening. The recorded medical history will be updated, if necessary, at admission to treatment period 1. Investigators should document the occurrence, signs, and symptoms of the participant's preexisting conditions, including all prior significant illnesses. Medical history will include alcohol consumption and smoking history, if applicable.

Illnesses first occurring or detected during the study and/or worsening of a concomitant illness during the study are to be documented as AEs in the eCRF in accordance with Section 12.5. All changes that are not present at baseline or described in the medical history and identified as clinically noteworthy must be recorded as AEs.

### 9.1.4. Eligibility Review

Participant eligibility will be reviewed per the inclusion criteria (Section 7.1) and exclusion criteria (Section 7.2) at the timepoints specified in the schedule of assessments (Table 3). Before randomization on Day 1, the eligibility review must be completed.

#### 9.1.5. Drug and Alcohol Screening

A urine drug test for prohibited substances, using a rapid, one-step screening test for simultaneous, qualitative detection of multiple drugs and drug metabolites will be performed at the timepoints specified in the schedule of assessments (Table 3). Results must be negative for study eligibility. However, if a participant has a positive result for a medically indicated substance such as benzodiazepines, and the Investigator determines that the participant was not abusing the substance, the positive result will not be exclusionary, provided that the Investigator consults with the Medical Monitor before enrolling or randomizing/dosing the participant.

An alcohol breath test using a portable breath alcohol measuring device will be performed. The test will be performed at screening, at admission to each treatment period and at random. If any of these tests are positive, the subject will not be allowed further participation in the study.

### 9.1.6. Serology Testing

Serum testing for HBsAg, IgM anti-HBc, HCV, and HIV will be performed at the timepoints specified in the schedule of assessments (Table 3).

### 9.1.7. Prior and Concomitant Medication

Any medication or therapy other than NKF-INS(A), US-NovoLog® and EU-NovoRapid® is considered concomitant medication (see Section 8.6.1) and should be recorded in the eCRF.

Relevant prior concomitant medication given within 3 weeks before screening and all medication given from screening until the EOS visit (within 2-11 days after last administration of the study drug) must be recorded.

All previous and on study COVID-19 vaccinations should be recorded in the eCRF.

#### 9.1.8. Other Screening Assessments

Other screening assessments include physical examination, height and weight, vital signs, 12-lead ECG, and safety laboratory assessments.

An oral glucose tolerance test will be conducted per site SOP. Oral glucose tolerance test may be completed after all other eligibility has been determined. For participants who re-screen, oral glucose tolerance test does not need to be repeated if completed within the last 6 months.

These assessments are also conducted at other timepoints as detailed in the schedule of assessments (Table 3).

### 10. PHARMACOKINETICS

# 10.1. Pharmacokinetic Sampling

#### 10.1.1. Blood Samples

Blood samples for PK analysis of NKF-INS(A), US-NovoLog® and EU-NovoRapid® will be collected at the timepoints indicated in Table 4. The actual date and time of each blood sample collection will be recorded. Actual time will be used for derivation of PK parameters.

Details of PK blood sample collection, processing, storage, and shipping procedures are provided in a separate laboratory manual.

#### 10.1.2. Pharmacokinetic Evaluation

The PK parameters will be derived for NKF-INS(A), US-NovoLog® and EU-NovoRapid® from serum concentrations by a validated PK analysis platform using standard noncompartmental methods (where data allow). A description of the PK parameters is provided in Table 5. A complete list of PK parameters will be provided in the statistical analysis plan (SAP).

**Table 5 Pharmacokinetic Parameters** 

| PK Parameter | Description |
|---|---|
| AUC <sub>0-4h</sub> | concentration-time curve from 0 to 4 hours |
| AUC <sub>0-6h</sub> | concentration-time curve from 0 to 6 hours |
| AUC <sub>6-12h</sub> | concentration-time curve from 6 to 12 hours |
| AUC <sub>0-12h</sub> | concentration-time curve from 0 to 12 hours/end of clamp |
| AUC <sub>0-t</sub> | concentration-time curve from 0 hour to the last quantifiable concentration |
| | time |
| $\mathrm{AUC}_{0\text{-}\infty}$ | concentration-time curve from 0 hour to infinity |
| $T_{\text{max}}$ | time to maximum serum concentration |
| $C_{max}$ | maximum observed insulin aspart concentration |
| t50%-early | time to half-maximum before C <sub>max</sub> |
| t50%-late | time to half-maximum after C <sub>max</sub> |
| t <sub>1/2</sub> | terminal elimination half-life |

PK parameters will be estimated using noncompartmental methods. Estimates of PK parameters will be listed and summarized (N, arithmetic and geometric mean, standard deviation [SD], coefficient of variation [CV%], median, minimum, and maximum) by treatment group), descriptively and graphically. The full analysis will be described in the prospective SAP that will be finalized prior to database lock.

# 10.2. Pharmacokinetic Analytical Methodology

The concentration of NKF-INS(A), US-NovoLog® and EU-NovoRapid® will be determined from the serum samples using a validated analytical method. Details of the method validation and sample analysis will be included with the final clinical study report.

### 11. PHARMACODYNAMICS

# 11.1. Pharmacodynamic Sampling

### 11.1.1. Blood Samples

Blood samples for NKF-INS(A), US-NovoLog<sup>®</sup>, and EU-NovoRapid<sup>®</sup> in serum will be collected at the timepoints indicated in the sample schedule shown in Table 4. The actual date and time of each blood sample collection will be recorded. Actual time will be used for derivation of PD parameters.

Details of PD blood sample collection, processing, storage, and shipping procedures are provided in a separate laboratory manual.

### 11.1.2. Pharmacodynamic Evaluation

The following PD parameters will be derived for NKF-INS(A), EU-NovoRapid<sup>®</sup>, and US-NovoLog<sup>®</sup> from serum concentrations by a validated PK analysis program using standard noncompartmental methods (where data allow):

The PD similarity will be assessed using the parameters provided in Table 6, and by assessing:

- Time from study drug administration until the blood glucose concentration has decreased by at least 5 mg/dL from baseline (onset of action)
- The difference between tGIR,50%-late and the onset of action (duration of action)
- Total amount of glucose infused during clamp procedure (Gtot)

A complete list of PD parameters will be provided in the SAP.

 Table 6
 Pharmacodynamic Parameters

| PD Parameter | Description |
|---|---|
| AUCGIR <sub>0-12h</sub> | Area under the GIR-time curve from 0 to 12 hours |
| GIR <sub>max</sub> | The maximum GIR of glucose |
| AUCGIR <sub>0-4h</sub> | Area under the GIR-time curve from 0 to 4 hours |
| AUCGIR <sub>0-6h</sub> | Area under the GIR-time curve from 0 to 6 hours |
| AUCGIR <sub>6-last</sub> | Area under the GIR-time curve from 6 hours until the end of clamp |
| AUCGIR <sub>0-t</sub> | Area under the GIR-time curve from 0 hours to the last quantifiable concentration time |
| $AUCGIR_{0-\infty}$ | Area under the GIR-time curve from 0 hours to the last quantifiable concentration time with extrapolation to infinity |
| AUCGIR <sub>0-end of clamp</sub> | Area under the GIR-time curve from 0 hours to end of clamp |
| T <sub>max</sub> .GIR | Time to maximum GIR |
| tGIR,50%-early | Time to half-maximum GIR before GIRmax |
| tGIR,50%-late | Time to half-maximum GIRe after GIR <sub>max</sub> (indicator of end of duration of action) |

Abbreviation: GIR = glucose infusion rate

Estimates of PD parameters will be listed and summarized (N, arithmetic and geometric mean, SD, CV%, median, minimum, and maximum) by treatment group, descriptively and graphically.

Endogenous insulin suppression via C-peptide measurements will also be explored. These values include corrected and uncorrected C-peptide concentrations. C-peptide corrected estimates of exogenous insulin will be calculated using Owen's method (Plum-Mörschel, 2022). If terminal phase of serum concentration-time profile has sufficient data points, apparent terminal elimination half-life ( $t\frac{1}{2}$ .z), apparent terminal elimination rate constant ( $\lambda$ z), mean residence time (MRT), clearance (CL/F), and volume of distribution (V/F) will be calculated.

### 11.1.3. Pharmacodynamic Analytical Methodology

The concentration of C-peptide, NKF-INS(A), US-NovoLog® and EU-NovoRapid® will be determined from the serum samples using a validated analytical method. Details of the method validation and sample analysis will be included with the final clinical study report.

#### 12. SAFETY ASSESSMENTS

Safety assessments (vital signs, physical examinations, ECG recordings, clinical laboratory assessments [hematology, clinical chemistry (including glucose), coagulation, and urinalysis], AE monitoring [including injection site reactions]) are to be performed as outlined in the schedule of assessments (Table 3).

## 12.1. Vital Signs

Vital signs (heart rate, respiratory rate, systolic and diastolic blood pressure, and temporal or ear temperature measurements) will be evaluated at the timepoints indicated in the schedule of assessments (Table 3). All vital signs will be measured after the participant has been resting in a supine position for at least 5 minutes. Height (without shoes) will be recorded at screening. Weight will be recorded at screening and on Day -1.

Vital sign measurements will be repeated if clinically significant abnormal or machine/equipment errors occur. Out-of-range blood pressure, respiratory rate, or heart rate measurements will be repeated at the Investigator's discretion. Any confirmed, clinically significant abnormal vital sign measurements must be recorded as AEs.

## 12.2. Physical Examination

A complete physical examination will be performed at screening (Visit 1). Physical examinations will be performed by a physician.

A full physical examination will include the following: evaluation for jaundice, pallor (anemia), cyanosis, clubbing, edema and lymphadenopathy; skin evaluation; fundoscopy; ear, nose and throat; cardiovascular assessment; respiratory assessment; abdominal evaluation; musculoskeletal assessment; neurological assessment. Other evaluations may be performed as deemed necessary by the Investigator.

A limited physical or symptom-driven examination to verify continued participant eligibility and to follow up regarding any change in medical history will be performed at the timepoints indicated in the schedule of assessments (Table 3) or at the Investigator's discretion. Symptom-driven, limited physical examinations may be performed as clinically indicated or at the discretion of the Investigator at any study visit. Clinically significant findings must be recorded as AEs.

# 12.3. Electrocardiograms

A 12-lead, resting ECG will be obtained at the timepoints indicated in the schedule of assessments (Table 3). ECG should always be performed after the participant has been resting in a supine position for at least 5 minutes.

At screening, the Investigator will examine the ECG traces for signs of cardiac disease that could exclude the participant from the study. An assessment of normal, clinically significant, or abnormal not clinically significant will be recorded; if the ECG is considered abnormal, the abnormality will be documented in the eCRF. ECGs will be repeated if clinically significant abnormalities are observed, or artifacts are present. Any confirmed, clinically significant abnormal ECG findings must be recorded as AEs.

### 12.4. Laboratory Assessments

Laboratory assessment samples (Table 7) are to be obtained at designated timepoints as detailed in the schedule of assessments (Table 3).

 Table 7
 Laboratory Assessments

| Hematology: | Clinical Chemistry: | Urinalysis (Dipstick): |
|---|---|---|
| Full and differential blood count | Alanine aminotransferase | Appearance |
| Hematocrit | Albumin | Glucose |
| Hemoglobin | Alkaline phosphatase | Blood |
| Mean corpuscular hemoglobin | Aspartate aminotransferase | Leucocytes |
| Mean corpuscular hemoglobin | Bilirubin (direct and total) | Ketone bodies |
| concentration | Urea | pН |
| Mean corpuscular volume | Creatine kinase* | Protein |
| Platelet count | Creatinine | Specific gravity |
| Red blood cell count | Electrolytes (calcium, chloride, | Urobilinogen |
| White blood cell count with | phosphorus, potassium, | Bilirubin |
| Differential (absolute values): | sodium) | Nitrite |
| Basophils | Gamma-glutamyl transferase | |
| Eosinophils | Glucose | |
| Lymphocytes | Lactate dehydrogenase | |
| Monocytes | Total cholesterol | |
| Neutrophils | Triglycerides | |
| | Oral glucose tolerance test | |
| Coagulation: | Other: | Serology: |
| PT | Urine drug | HBsAg |
| aPTT | Human insulin antibodies | IgM anti-HBc |
| INR | | HCV |
| | | HIV |

Abbreviations: anti-HBc = hepatitis B core antigen; aPTT = activated partial thromboplastin time; CK-MB = creatine kinase MB; HBsAg = hepatitis B surface antigen; HCV = hepatitis C virus; HIV = human immunodeficiency virus; IgM = immunoglobulin M; INR = international normalized ratio; PT = prothrombin time.

Vitamin D retest is allowed once.

The tests detailed in Table 7 will be performed. All laboratory reports must be reviewed, signed, and dated by the Investigator. A legible copy of all reports must be filed with the participant's medical record (source document) for that visit. Any laboratory test result considered by the Investigator to be clinically significant should be considered an AE (clinically significant AEs include those that require an intervention). Clinically significant abnormal values occurring during the study will be followed up until repeat test results return to normal, stabilize, or are no longer clinically significant.

Further laboratory assessments outside the protocol-defined schedule may be obtained at the discretion of the Investigator and used for other clinical treatment decisions.

### 12.5. Injection Site Assessment

The injection site and surrounding area will be assessed by the investigator at 1 min and 15 min post-dose on Day 1 and at the EOS visit. Reactions to the study drug injection will be documented using a numerical scoring system.

<sup>\*</sup> In case of elevated creatine kinase, CK-MB may be performed, at the discretion of the Investigator

#### **12.6.** Adverse Events

#### 12.6.1. Definitions

#### **12.6.1.1.** Adverse Event

Any untoward medical occurrence in a patient or clinical investigation subject administered an investigational product which does not necessarily have to have a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product.

#### 12.6.1.2. Adverse Reaction

A response to a medicine in humans which is noxious and unintended, and which occurs at any dose, and which can also result from overdose, misuse, or abuse of a medicine. Response to a medicinal product in this context means that a causal relationship between the medicinal product and an AE is at least a reasonable possibility.

#### 12.6.1.3. Serious Adverse Event

Any untoward medical occurrence, in the view of either the Investigator or Sponsor, that:

- Results in death
- Is life-threatening
  - An AE is life-threatening if the participant was at immediate risk of death from the event as it occurred (i.e., it does not include a reaction that might have caused death if it had occurred in a more serious form).
- Requires or prolongs inpatient hospitalization
  - A hospitalization is defined as ≥24 hours in hospital or an overnight stay. Complications occurring during hospitalization are AEs and SAEs if they cause prolongation of the current hospitalization. Hospitalization for elective treatment of a preexisting, non-worsening condition is not, however, considered an AE. The details of such hospitalizations must be recorded in the medical history/procedures or physical examination page of the eCRF.
- Results in persistent or significant disability/incapacity
  - An AE is incapacitating or disabling if it results in a substantial and/or permanent disruption of the participant's ability to carry out normal life functions.
- Results in a congenital anomaly/birth defect
- Is another medically important event

In addition, medical and scientific judgment is required to decide if prompt notification is required in situations other than those defined for SAEs. This may include any event that the Investigator regards as serious that did not strictly meet the criteria above but may have jeopardized the participant or required intervention to prevent one of the outcomes listed

above, or that would suggest any significant hazard, contraindication, AE, or precaution that may be associated with the use of the study treatment.

Other important medical events that may not be immediately life-threatening or result in death or hospitalization, based upon appropriate medical judgment, are considered SAEs if they are thought to jeopardize the participant and/or require medical or surgical intervention to prevent one of the outcomes defining an SAE. SAEs are critically important for the identification of significant safety problems; therefore, it is important to consider both the Investigator's and the Sponsor's assessment.

#### 12.6.1.4. Pre-treatment Adverse Event

An AE with a start date and time before the first dose of study drug.

#### 12.6.1.5. Treatment-Emergent Adverse Event

An AE with a start date and time on or after the first dose of study drug.

### 12.6.1.6. Unexpected Adverse Reaction

An adverse reaction in which the nature, specificity, severity, and outcome is not consistent with the referenced safety information.

#### 12.6.2. Adverse Event Collection, Assessment and Reporting

#### 12.6.2.1. Observation Period for Assessment of Adverse Events

For the purposes of this study, the period of observation for collection of AEs (including nonserious AEs and SAEs) extends from the time the participant begins study treatment (Day 1) until the EOS visit (within 2-11 days after last administration of the study drug). If a participant withdraws or is discontinued from the study by the Investigator, AEs should be collected from the time the participant begins study treatment (Day 1) up to the completion of EOS assessments.

#### 12.6.2.2. Parameters for Adverse Events Collection

All nonserious AEs and SAEs will be recorded on the AE eCRF. SAEs will also be immediately reported to the Sponsor safety representative in accordance with Section 12.5.5.

Nonserious and SAEs will be documented in the clinical database with the highest severity documented during the duration of each serious or nonserious episode. Each AE is to be documented in the eCRF with reference to date of onset, severity, relationship to study drug, treatment of event, and outcome.

All AEs are to be followed up until resolution or a stable clinical endpoint is reached, as determined by the Investigator. Changes in AEs and resolution dates are to be documented in the eCRF.

Participants will be instructed by the Investigator to report AEs at each study visit. All volunteered, elicited, and observed AEs are to be recorded. A consistent methodology of nondirective questioning should be adopted for eliciting AE information at all participant evaluation timepoints. Examples of nondirective questions include the following:

- "How are you feeling?"
- "How have you felt since your last clinic visit?"

- "Have you had any new or changed health problems since you were last here?"
- "Have you taken any new medications since your last visit?"

The following considerations should also be made regarding AE and SAE reporting:

- All medical and psychiatric conditions present at screening (i.e., conditions present before the AE reporting period) will be considered preexisting conditions and documented in the medical history eCRF. A preexisting condition is not to be reported as an AE. If a preexisting condition worsens during the study treatment period, the event should be reported as an AE. Planned hospitalization for a preexisting condition, or a procedure required by the protocol, without serious deterioration in health, is not considered an SAE.
- Diagnostic and therapeutic noninvasive and invasive procedures, such as surgery, should not be reported as AEs. A medical condition for which an unscheduled procedure was performed, should however be reported if it meets the definition of an AE. For example, an acute appendicitis, and not the appendectomy, should be reported as the AE.
- Clinically significant abnormal laboratory findings (e.g., hematology, clinical chemistry [including glucose], coagulation, and urinalysis) or other abnormal assessments (e.g., in ECG results and vital signs), meeting the definition of an AE or SAE, that are detected during the study or are present at baseline and significantly worsen following the start of the study will be reported as AEs or SAEs. The Investigator will exercise his/her medical and scientific judgment in deciding whether an abnormal laboratory finding, or other abnormal assessment is clinically significant.

Special situations are non-standard medical conditions that provide valuable information (e.g., clinical, safety) about a medicinal product, even when special situations do not occur in association with an AE or medical condition. Special situations, defined in this protocol as events of accidental overdose, medication error, and drug misuse, are not in and of themselves AEs but may result in AEs. Each AE associated with a special situation should be recorded in the AE eCRF. If the associated AE fulfills seriousness criteria, the event should be reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event).

In the event of an accidental overdose, medication error or drug misuse special situation, the Investigator should:

- Inform the Medical Monitor immediately.
- Closely monitor the participant for an AE/SAE and laboratory abnormalities.
- In the event of an accidental overdose: document the quantity of excess dose in the eCRF.

#### 12.6.3. Assessment of Event Severity

The Investigator will use the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 to describe the severity of AEs. AEs not listed in the CTCAE will be graded as follows:

| 11111 1115(11) | Version 2.0 |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Self-care ADL refers to bathing, dressing & undressing, feeding self, using the toilet, taking medications, and not bedridden. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to the AE. |

## 12.6.4. Relationship to Study Treatment

Specific guidelines for classifying AEs by relationship to study treatment are given in Table 8.

### Table 8 Classification of Adverse Events by Relationship to Study Treatment

**NOT RELATED:** There is not a reasonable possibility that the administration of the study intervention caused the event, there is no temporal relationship between the study intervention and event onset, or an alternate etiology has been established.

**RELATED:** The AE is known to occur with the study intervention, there is a reasonable possibility that the study intervention caused the AE, or there is a temporal relationship between the study intervention and event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study intervention and the AE.

#### 12.6.5. Serious Adverse Event Reporting

Any SAE occurring during the course of the study within the defined AE reporting window, must be immediately reported to the appropriate Sponsor safety representative (PrimeVigilance) within 1 calendar day (i.e., within 24 hours) of the investigational site's initial awareness of the event. The study SAE Report Form, provided by the Sponsor, will be utilized for reporting safety information to the Sponsor safety representative and completed in English. For fatal or life-threatening treatment-emergent SAEs, where important or relevant information is missing, active follow up will be undertaken immediately by the Investigator.

A post-study AE or SAE is defined as any event that occurs outside of the AE/SAE monitoring period. Investigators are not obligated to actively monitor AEs or SAEs of such study participants. However, if the Investigator learns of any AE or SAE, including a death, at any time after a participant has completed the study, and it is considered reasonably related to the study treatment, the Investigator should promptly notify the Sponsor safety representative within 24 hours of becoming aware of the event.

Investigators or other site personnel will inform the Sponsor safety representative of any follow-up information on a previously reported SAE within 1 calendar day (i.e., within 24 hours) of the investigational site's awareness of the new information. All SAEs will be followed until satisfactory resolution, until the Investigator deems the event to be chronic, or

the participant is stable. Other supporting documentation of the event may be requested by the Sponsor or Sponsor safety representative and should be provided by the Investigator as soon as possible.

The Sponsor will notify regulatory authorities and participating Investigators of any reportable SAEs for NKF-INS(A), US-NovoLog<sup>®</sup>, and EU-NovoRapid<sup>®</sup>) in an expedited fashion in accordance with local requirements. Where required and in accordance with local requirements, the Sponsor will ensure unblinding of subject treatment assignment for the purposes of reporting the event to regulatory authorities. IRBs/IECs will be promptly notified, in accordance with local regulations, of all reportable SAEs involving risk to human participants. Where reportable SAEs are identified for referenced products, i.e., US-NovoLog<sup>®</sup> and EU-NovoRapid<sup>®</sup>, the Sponsor will ensure the product manufacturer is notified within the same expedited timelines as regulatory authorities.

For further guidance on the definition of an SAE, see Section 12.5.1.3.

# 12.7. Drug-Induced Liver Injury Monitoring

For new elevations in transaminases greater than 2 × the upper limit of normal (ULN) in participants with normal baseline values, repeat measurement will be performed within 48 hours. If elevations persist, participants will be evaluated for other causes of transaminase elevations and with tests of hepatic function. If no other cause is found, then the participants will be monitored closely and the drug discontinued as per the recommendations in the FDA Guidance for Industry – Drug-Induced Liver Injury: Premarketing Clinical Evaluation (US FDA, 2009).

The participant should be followed until resolution of symptoms or signs in the following situations:

- Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >8 × ULN.
- ALT or AST >5 × ULN for more than 4 days during the 7-day treatment period.
- ALT or AST >3 × ULN (and total bilirubin >2 × ULN or international normalized ratio [INR] >1.5).
- ALT or AST >3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).

#### 12.7.1. Pregnancy

After administration of study treatment, any known cases of pregnancy in female partners of male study participants will be reported until the male participant completes or withdraws from the study and within 90 days of their exposure to study treatment. The Investigator may arrange counseling for pregnant female partners of male study participants by a specialist to discuss the risks of continuing with the pregnancy and the possible effects on the fetus. The pregnancy will be reported immediately by faxing/emailing a completed pregnancy report to the Sponsor safety representative (or designee) within 24 hours of knowledge of the event. The pregnancy will not be processed as an AE/SAE; however, the Investigator must follow up with female partners of male study participants until completion of the pregnancy, and must assess the outcome in the shortest possible time, but not more than 30 days, after completion of the pregnancy. The Investigator should notify the Sponsor (or designee) of the pregnancy outcome by submitting a follow-up pregnancy report. If the outcome of the pregnancy involved spontaneous or therapeutic abortion (any congenital anomaly detected in

an aborted fetus is to be documented as an SAE), stillbirth, neonatal death, or congenital anomaly, the Investigator will report the SAE by faxing/emailing a completed pregnancy report form to the Sponsor safety representative (or designee) within 24 hours of knowledge of the event. Any pregnancy in female partners of male study participants will be followed to term, and the status of the mother and child will be reported to the Sponsor after delivery.

Contraception guidance is provided in Appendix 1.

#### 12.7.2. Accidental Overdose, Medication Error, or Drug Misuse

Accidental overdose, medication error, and drug misuse, hereafter collectively referred to as "special situations," are defined as follows:

- Accidental overdose: accidental administration of a drug in a quantity that is higher than the assigned dose.
- Medication error: accidental deviation in the administration of a drug. In some cases, a medication error may be intercepted before administration of the drug.
- Drug misuse: intentional deviation in the administration of a drug that does not qualify as drug abuse.

Cases of accidental overdose, drug misuse, or medication error without manifested signs or symptoms are not considered AEs. Adverse events associated with an overdose will be documented according to Section 12.5.5. SAEs associated with overdose should be reported according to the procedure outlined in Section 12.6.2. All cases of overdose (with or without associated AEs) will be documented on the eCRF.

### 13. OTHER ASSESSMENTS

# 13.1. Euglycemic Clamp Procedure

NKF-INS(A), US-NovoLog® and EU-NovoRapid® will be administered using a euglycemic glucose clamp at targeted blood glucose concentrations. The euglycemic glucose clamp will be conducted using a manual clamp technique, which will continuously monitor the subject's blood glucose and administer GIR to maintain blood glucose close to the target blood glucose concentration. The clamp procedure will be initiated, maintained, and terminated, in accordance with the site SOPs. The participant's blood glucose will be maintained within a pre-defined target window per site SOP and clinical judgment for the participant by manually adjusting the GIR.

Blood samples will be collected at pre-specified intervals before and up to 12 hours after dosing for measurement of blood glucose, serum insulin, and C-peptide as shown in the schedule of assessments (Table 3).

#### 14. STATISTICAL ANALYSIS

An SAP will be prepared after the protocol is approved. The SAP will provide further details regarding the definition of analysis variables and analysis methodology to address all study objectives. The SAP will serve as a complement to the protocol and supersedes it in case of differences.

The statistical evaluation will be performed using R version 4.0 or higher. All data will be listed, and summary tables and figures will be provided. Summary statistics will be presented by treatment group, to the extent possible. For continuous variables, data will be summarized with the number of participants (N), arithmetic mean, SD, median, minimum, and maximum by treatment group. Geometric mean and CV% will be presented as appropriate, by treatment group. For categorical variables, data will be tabulated with the number and proportion of participants for each category by treatment group.

# **14.1.** Determination of Sample Size

A literature review of similar studies was conducted in order to inform the assumptions for the sample size, for the primary endpoints of  $AUC_{0-\infty}$  and  $C_{max}$  (see Table 9).

 Table 9.
 Studies Referenced for Sample Size Assumptions

| Program | AUC <sub>0-t</sub> | AUC₀-∞ | C <sub>max</sub> | GIR <sub>max</sub> | AUCGIR | Median | Sample<br>Size |
|---|---|---|---|---|---|---|---|
| Innovator<br>[NovoLog<br>USPI] | | 9.8% | 25.30% | 18.0% | 17.6% | | 24 |
| Mylan (HV)<br>[Hovelmann,<br>2021] | 32.0% | 32.0% | 30.90% | 18.5% | 17.5% | | 71 |
| Sanofi (T1DM)<br>[Kapitza, 2020] | 16.0% | 15.7% | 30.75% | 30.8% | 30.0% | | 30 |
| Yichang HEC<br>Changjiang<br>Pharmaceutical<br>Co., Ltd (HV)<br>[Liu, 2021] | 17.0% | 16.5% | 31.0% | 22.0% | 27.0% | | 30 |
| Mean | 21.7% | 18.5% | 29.5% | 22.3% | 23.0% | 22.3% | |
| Median | 17.0% | 16.1% | 30.8% | 20.3% | 22.3% | | |

Abbreviation: GIR = glucose infusion rate; HV = healthy volunteers; T1DM = type 1 diabetes mellites

The CV value ranged from 23.8% to 30.8%, with a mean value of 25.4%. The CV of the Innovator study was 25.3%. Based on the above data, the CV value is selected as 26%.

The sample size is calculated using PASS software with following parameters including 90% power, drop rate 20%,  $\alpha$ =0.05, 90% confidence interval (CI), assumed actual ratio 0.95 within 80-125%, N=40; taking account of 20% dropout, the sample size is determined as N=54 to have at least 36 evaluable participants.

# 14.2. Analysis Populations

The following analysis populations are planned for this study:

### **Screening Population**

All individuals who provide informed consent and provide demographic and/or baseline screening assessments, regardless of the participant's randomization status.

### **Enrolled Population**

The Enrolled Population will include all individuals who sign the ICF.

### Safety Population

The Safety Population will include all participants who receive any amount of study treatment. This population will be used for the analysis of safety.

### Pharmacokinetic Concentration Population

The PK Concentration Population will include all participants in the Safety Population who received any amount of study treatment and have at least 1 post-baseline reportable PK result.

### Pharmacokinetic Parameter Population

The PK Parameter Population will include all participants in the PK Concentration Population who have at least 1 PK parameter derived.

### Pharmacodynamic Parameter Population

The PD Parameter Population will include all participants in the Safety Population who have at least 1 PD parameter derived.

# 14.3. Pharmacokinetic Analysis

The primary PK objective is to compare the PK of NKF-INS(A) to US-approved and EU-authorized insulin aspart to demonstrate PK similarity for insulin aspart. The secondary PK objective is to evaluate additional PK parameters of NKF-INS(A) compared to US-approved and EU-authorized insulin aspart. Details on the endpoints are provided in Table 1.

PK concentrations and parameter data will be listed and summarized descriptively (N, arithmetic and geometric mean, SD, CV%, median, minimum, and maximum) by treatment group and graphically.

Biosimilarity between the test product and the US-approved and EU-authorized insulin aspart will be considered separately, i.e., test product vs US-approved product and test product vs EU-authorized product. Biosimilarity of the test and reference products will be assessed on the basis of the 90% Cis for estimates of the geometric mean ratios between the primary PK parameters of the test and reference products in relation to the conventional bioequivalence range of 80% to 125%. The test product will be compared to the reference product by means of statistical analysis with respect to the primary PK parameters using an analysis of variance after logarithmic transformation of the data. Point estimates and 90% Cis for the "test/reference" geometric mean ratios of these parameters will be provided. The primary PK parameters that will be used for the bioequivalence assessment are  $C_{max}$  and  $AUC_{0-t}$ . All other PK-related assessments of equivalence will be considered secondary.

Any missing samples or non-reportable concentration values will be disregarded in the PK analysis.

Refer to the SAP for full details.

## 14.4. Pharmacodynamic Analysis

The primary PD objective is to compare the PD of NKF-INS(A) to US-approved and EU-authorized insulin aspart injection by examining GIR profiles after a single SC dose. The secondary PD objective is to evaluate the additional parameters NKF-INS(A) compared to US-approved and EU-authorized insulin aspart. Details on the endpoints are provided in Table 1. PD concentrations and parameter data will be listed and summarized descriptively (N, arithmetic and geometric mean, SD, CV%, median, minimum, and maximum) by treatment group and graphically.

As for PK similarity, biosimilarity between the test product and the US-approved and EU-authorized insulin aspart will be considered separately, i.e., test product vs US-approved product and test product vs EU-authorized product. Biosimilarity of the test and reference products will be assessed on the basis of the 95% Cis for estimates of the geometric mean ratios between the primary PK parameters of the test and reference products in relation to the conventional bioequivalence range of 80% to 125%. The test product will be compared to the reference product by means of statistical analysis with respect to the primary PD parameters using an analysis of variance after logarithmic transformation of the data. Point estimates and 90% and 95% Cis for the "test/reference" geometric mean ratios of these parameters will be provided. The primary PD parameters that will be used for the bioequivalence assessment are GIR<sub>max</sub> and AUCGIR<sub>0-t</sub>. All other PD-related assessments of equivalence will be considered secondary.

All PD analyses will be based on the PD Parameter Population. Refer to the SAP for full details.

## 14.5. Safety Analysis

All analyses of safety will be conducted on the Safety Population unless otherwise specified in the SAP.

All reported AEs will be graded using NCI CTCAE version 5.0 and will be coded using the Medical Dictionary for Regulatory Activities, version 26.0. The incidence of treatment-emergent AEs (TEAEs) will be included in incidence tables. Events with missing onset dates will be included as treatment-emergent. If a participant experiences more than 1 occurrence of the same AE, the occurrence with the greatest severity and the closest association with the study treatment will be used in the summary tables. All TEAEs will be summarized by treatment group (NKF-INS(A), US-NovoLog<sup>®</sup>, and EU-NovoRapid<sup>®</sup>) as follows:

- All AEs
- Grade ≥3 AEs
- AEs related to study treatment, including related Grade  $\geq$ 3 AEs
- All adverse reactions
- SAEs

All AEs will be listed by participant, along with information regarding onset, duration, relationship and severity to study treatment, action taken with study treatment, treatment of event, and outcome.

Clinical laboratory data (hematology, clinical chemistry [including glucose], coagulation, and urinalysis) and vital signs (heart rate, respiratory rate, systolic and diastolic blood pressure, and temporal or ear temperature measurements) will be summarized by treatment group and

scheduled visits using descriptive statistics, including mean values and mean change from screening values, as well as numbers of participants with values outside limits of the normal range at each timepoint. Shift tables will be provided presenting change from screening values to the last EOS visit.

The frequency of ECG abnormalities (e.g., heart rate, PR interval, QRS complex, and QT-interval corrected by Fridericia's formula [Fridericia's corrected QT]) will be summarized by treatment group and scheduled visits using counts and percentages.

Participant ECG status (normal, abnormal clinically significant, or abnormal not clinically significant) may be summarized for each scheduled ECG and shifts from screening may be tabulated.

Injection site reactions will be summarized by treatment group and scheduled visits. The number and percentage of participants having reactions at each assessment timepoint, overall and by specific reaction subtype, will be presented.

Summary tables will be provided for concomitant medications initiated during the study period.

Clinically significant changes in physical examination findings and laboratory abnormalities will be listed as AEs.

# 14.6. Other Analyses

All other safety variables will be listed.

## 14.7. Interim Analysis

No interim analysis is planned.

## 14.8. Data Monitoring Committee

Not applicable.

#### 15. STUDY MANAGEMENT

## **15.1.** Approval and Consent

### 15.1.1. Compliance with Laws and Regulations

This study will be conducted in full conformance with the ICH E6 guideline for GCP and the principles of the Declaration of Helsinki or all relevant laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual.

The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the EU or European Economic Area will comply with the EU Clinical Trial Regulation (CTR).

## 15.1.2. Institutional Review Board/Independent Ethics Committee

This protocol, protocol amendments (if applicable), Investigator's Brochure, the ICFs, recruitment material and participant information sheets, any information to be given to the participant, and relevant supporting information must be submitted to the IEC/IRB by the Principal Investigator (PI) and reviewed and approved by the IEC/IRB before the study is initiated; no participant may undergo any procedure for determining eligibility for this study until IEC/IRB approval is obtained.

The PI is responsible for providing written summaries of the status of the study to the IEC/IRB annually or more frequently in accordance with the requirements, policies, and procedures established by the IEC/IRB. Investigators are also responsible for promptly informing the IEC/IRB of any protocol amendments. The PI must receive approval/acknowledgement from the IEC/IRB before implementation of the amendment.

In addition to the requirements for reporting all AEs to the Sponsor, Investigators must comply with requirements for reporting SAEs to the local health authority and IEC/IRB.

Investigators may receive written investigational new drug safety reports or other safety-related communications from the Sponsor. Investigators are responsible for ensuring that such reports are reviewed and processed in accordance with health authority requirements and the policies and procedures established by their IEC/IRB and archived in the site's study file.

#### 15.1.3. Informed Consent Process

#### 15.1.3.1. Consent and Other Informational Documents Provided to Participants

Consent forms describing in detail the study intervention, study procedures, and risks are given to the participant and written documentation of informed consent is required before protocol-specific procedures are performed.

#### 15.1.3.2. Consent Procedures and Documentation

Informed consent is a process that is initiated before the participant's agreeing to participate in the study and continues throughout the study participation. Consent forms will be IRB-approved, and the participant will be asked to read and review the document. The Investigator will explain the research study to the participant and answer any questions that may arise. A verbal explanation will be provided in terms suited to the participant's comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participants. Participants will have the opportunity to carefully review the written

consent form and ask questions before signing. The participants should have the opportunity to discuss the study with their family or surrogates or think about it before agreeing to participate. The participant will sign the informed consent document before any procedures being done specifically for the study. Participants must be informed that participation is voluntary and that they may withdraw from the study at any time, without prejudice. A copy of the informed consent document will be given to the participants for their records. The informed consent process will be conducted and documented in the source document (including the date), and the form signed, before the participant undergoes any study-specific procedures. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

## 15.2. Study Discontinuation and Closure

This study may be temporarily suspended or prematurely terminated at any time by the Sponsor, IEC/IRB and/or regulatory authorities if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the Sponsor to Investigators, the IRBs/IECs and regulatory authorities, as well as to any contract research organizations used in the study and provide the reason for termination. If the study is prematurely terminated or suspended, the PI will promptly inform study participants and the IRBs/IECs. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule.

## 15.3. Confidentiality and Privacy

Participant confidentiality and privacy are strictly held in trust by the participating Investigators, their staff, and the Sponsor. This confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study, or the data will be released to any unauthorized third party without prior written approval of the Sponsor.

All research activities will be conducted in as private a setting as possible.

The study monitor, other authorized representatives of the Sponsor, representatives of the IRB, regulatory agencies may inspect all documents and records required to be maintained by the Investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

The study participants' contact information will be securely stored at each CRU for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, institutional policies, or Sponsor requirements.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the data management company responsible for data management, analysis, and reporting. This will not include the participants' contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by CRUs and by data management research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived by the Sponsor.

All information generated in this study must be considered highly confidential and must not be disclosed to any people not directly concerned with the study without written prior permission from the Sponsor. Authorized regulatory officials and Sponsor personnel (or their representatives) will be allowed full access to inspect and copy the records. All study investigational products, participant bodily fluids, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by the Sponsor. Participants will only be identified by unique participant numbers in eCRFs.

Every participant will be given a copy of each version of the ICF that he signs before and during the study. Each ICF may also include authorization allowing the institution, Investigator, and Sponsor to use and disclose personal health information in compliance with the Health Insurance Portability and Accountability Act of 1996.

# 15.4. Future Use of Stored Specimens and Data

No future use of stored specimens is planned.

Once samples have been analyzed, specimens will be destroyed. If no analyses have been completed within 5 years following EOS, samples will be destroyed.

## 15.5. Safety Oversight

Safety oversight will be under the direction of the Medical Monitor in concert with the Sponsor Medical Director as outlined in the Safety Management Plan and Medical Monitoring Plan.

## 15.6. Clinical Monitoring

CRU monitoring is conducted to ensure that the rights and well-being of study participants are protected. Study monitors will perform ongoing source data verification to confirm that the reported study data are accurate, complete, and verifiable from source documents, and that the conduct of the study is in compliance with the currently approved protocol/amendment(s), with ICH GCP, and with applicable regulatory requirement(s).

Monitoring for this study will be performed by a Sponsor-contracted Contract Research Organization (CRO).

Details of CRU monitoring are documented in a Clinical Monitoring Plan (CMP). The CMP describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports.

Independent audits will be conducted by a Sponsor-designated, qualified person to ensure monitoring practices are performed consistently across all participating sites and that monitors are following the CMP.

# **15.7. Quality Assurance and Quality Control**

Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site for clarification/resolution.

Following written SOPs, the monitors will verify that the clinical study is conducted, data are generated, and biological specimens are collected, documented (recorded), and reported in

compliance with the protocol, ICH GCP, and applicable regulatory requirements (e.g., Good Laboratory Practices, Good Manufacturing Practices).

The investigational site will provide direct access to all study-related sites, source data/documents, and reports for the purpose of monitoring and auditing by the Sponsor, and inspection by local and regulatory authorities.

### 15.8. Data Handling and Record Keeping

### 15.8.1. Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical study staff at the CRU under the supervision of the site Investigator. The Investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

Data recorded in the eCRF derived from source documents should be consistent with the data recorded in the source documents.

Clinical data (including AEs, concomitant medications, and adverse reactions data) and clinical laboratory data will be entered into a 21 Code of Federal Regulations (CFR) Part 11-compliant data capture system provided by the CRO. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be entered directly from the source documents as outlined in the Case Report Form Completion Guidelines.

### 15.8.2. Study Records Retention

The Investigator shall retain and preserve a copy of all records and data generated in the course of the study, specifically those defined by ICH GCP E6 as essential until:

- A minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or
- A least 2 years have elapsed since the formal discontinuation of clinical development of the study drug.

These documents should be retained for a longer period, however, if required by local regulations or requested by the Sponsor. No records will be destroyed without the written consent of the Sponsor. It is the responsibility of the Sponsor to inform the Investigator when these documents no longer need to be retained.

At the end of the retention period, the Investigator shall notify the Sponsor in writing of her/his intent to destroy such material. The Sponsor shall have 30 days to respond to the Investigator's notice and shall have further opportunity to retain such materials.

#### 15.9. Protocol Amendment and Protocol Deviation

#### 15.9.1. Protocol Amendment

Amendments to the protocol that entail corrections of typographical errors, clarifications of confusing wording, changes in study personnel, and minor modifications that have no effect on the safety of participants, or the conduct of the study will be classed as administrative

amendments. The Sponsor will ensure that acknowledgement is received, filed, and submitted according to local regulations.

Amendments that are classed as substantial amendments must be submitted by the PI to the appropriate regulatory authorities and the IECs/IRBs for approval, and will not be implemented at sites until such approvals are received other than in the case of an urgent safety measure.

#### 15.9.2. Protocol Deviations

A protocol deviation is any noncompliance with the clinical study protocol, ICH GCP, or applicable SOPs and site manuals. In addition, the study will be conducted in accordance with the applicable regulatory requirements of the country where the study is being conducted. The noncompliance may be either on the part of the participant, the Investigator, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly.

It is the responsibility of the site Investigator to use continuous vigilance to identify and report deviations as soon as possible. All deviations must be addressed in study source documents and must be sent to the reviewing IRB/IEC, per their SOPs. The site Investigator is responsible for knowing and adhering to the reviewing IRB/IEC requirements. Further details about the handling of protocol deviations will be included in the Protocol Deviation Plan, Data and Medical Management Plans, and SAP.

The study will be conducted as described in this protocol, except for an emergency situation in which the protection, safety, and well-being of the participant requires immediate intervention, based on the judgment of the Investigator (or a responsible, appropriately trained professional designated by the Investigator). In the event of a significant deviation from the protocol due to an emergency, accident, or mistake, the Investigator (or designee) must contact the Medical Monitor and the Sponsor at the earliest possible time by telephone. This will allow an early joint decision regarding the participant's continuation in the study. This decision will be documented by the Investigator and the Medical Monitor.

### **15.10.** Ethical Considerations

This study will be conducted in accordance with this protocol, the accepted version of the Declaration of Helsinki and/or all relevant federal regulations, as set forth in Parts 50, 56, 312, Subpart D, of Title 21 of the CFR and EU 536/2014, Annex 1, D, 17 (a); and in compliance with ICH GCP guidelines, as well as local regulatory requirements in countries/regions where the study is being conducted.

IECs/IRBs will review and approve this protocol and the ICF. All participants are required to give written informed consent before participation in the study.

### 15.11. Financing and Insurance

Details on finance and insurance will be provided in a separate agreement between the Investigator and the Sponsor.

## **15.12.** Publication Policy

This study will be registered at ClinicalTrials.gov, and results information from this study will be submitted to ClinicalTrials.gov and local registries as required by local regulation.

Any publication proposed to be published by Investigator shall be provided to Sponsor prior to publication or other disclosure. Due regard shall be given to, and adjustments to publication content and timing shall be made, based upon Sponsor's legitimate interests in publication review, e.g., ensuring compliance with the statistical analyses for the primary endpoints of the study according to, and consistent with, the Protocol; identifying any inaccuracies or errors in data analyses; obtaining patent protection; coordinating and maintaining the proprietary nature of submissions to health authorities; and protection of Confidential Information. In order to ensure that all publications related to Sponsor studies are responsible, ethical, timely, legally compliant, and scientifically fair and balanced, all publications contemplated hereunder will follow prevailing industry guidelines for good publication practices, including, but not limited to guidelines published by the International Committee of Medical Journal Editors and the position statements and guidelines published by the International Society for Medical Publication Professionals regarding good publication practices

In the event that Institution or Investigator proposes to publish or otherwise disclose (whether orally or in writing) any findings, data, or results regarding the study, a draft thereof shall be submitted to Sponsor at least forty-five (45) days prior to submission for publication or other disclosure. Procedures set forth shall apply to publication of research and data derived from the study even when the study is terminated early or suspended for any reason. Results from the study shall not be made available to any third party by the Institution, Investigator, or any Study Site Team Participant outside of the publication procedures set out above.

## **15.13.** Conflict of Interest Policy

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual, perceived, or potential conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have an actual, perceived, or potential conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial. The study leadership has established policies and procedures for all study group members to disclose all actual, perceived, or potential conflicts of interest and will establish a mechanism for the management of all reported conflicts of interest.

#### 16. REFERENCES

Ampudia Blasco FJ. Biosimilars and novel insulins. Am J ther. 202;27(1):e52-e61.

Chen W, Lu J, Plum-Mörschel L, Andersen G, Zijlstra E, He A, et al. Pharmacokinetic and pharmacodynamic bioequivalence of Gan & Lee insulin analogues aspart (rapilin®), lispro (prandilin®) and glargine (basalin®) with EU- and US-sourced reference insulins. Diabetes Obes Metab. 2023;1-9.

Clinical Trial Facilitation Group. Recommendations related to contraception and pregnancy testing in clinical trials. 2014. Accessed at:

https://www.hma.eu/fileadmin/dateien/Human\_Medicines/01-About\_HMA/Working\_Groups/CTFG/2014\_09\_HMA\_CTFG\_Contraception.pdf

Drai RV, Karonova TL, Mayorov AY, Makarenko IE, Dorotenko AR, Kulesh VS, et al. Clinical pharmacology of insulin aspart biosimilar comparability in hyperinsulinemic euglycemic clamp procedure. Clinical Pharmacology in Drug Development. 2022;11(8):922-929

Heinemann L, Davies M, Home P, Forst T, Vilsbøll T, Schnell O. Understanding Biosimilar Insulins - Development, Manufacturing, and Clinical Trials. J Diabetes Sci Technol. 2023 Nov;17(6):1649-1661.

Hövelmann U, Raiter Y, Chullikana A, Liu M, Donnelly C, Lawrence T, et al. Pharmacokinetic and pharmacodynamic bioequivalence of biosimilar MYL-1601D with US and European insulin aspart in healthy volunteers: a randomized, double-blind, crossover, euglycaemic glucose clamp study. Diabetes Obes Metab. 2021;23:2670-2678.

Kapitza C, Nosek L, Schmider W, Teichert L, Nowotny I. Single-Dose Euglycemic Clamp Study Demonstrating Pharmacokinetic and Pharmacodynamic Similarity Between SAR341402 Insulin Aspart and US- and EU-Approved Versions of Insulin Aspart in Subjects with Type 1 Diabetes. Diabetes Technol Ther. 2020 Apr;22(4):278-284.

Liu H, Yu H, Sun L, Qiao J, Wan S, Li S, Li J, Tan H, Yu Y. Similar pharmacokinetics and pharmacodynamics of a new biosimilar and reference insulin aspart in healthy Chinese males. Sci Rep. 2021 May 4;11(1):9495.

NovoLog<sup>®</sup> (insulin aspart) United States Prescribing Information. 2023. Novo Nordisk Inc, DK-2880 Bagsvaerd, Denmark.

NovoRapid Summary of Product Characteristics. 2021. Novo Nordisk Limited, Gatwick, West Sussex, RH6 0PA, UK.

Plum-Mörschel L, Singh G, Murugesan SNM, Marwah A, Panda J, Loganathan S, et al. Pharmacokinetic and pharmacodynamic equivalence of Biocon's biosimilar insulin-R with the US-licensed Humulin<sup>®</sup> R formulation in healthy subjects: results from the RHINE-1 (Recombinant Human Insulin Equivalence-1) study. Diabetes Obes Metab. 2022;24:713-721.

World Health Organization. Coronavirus disease (COVID-19) pandemic. Accessed at: <a href="https://www.who.int/emergencies/diseases/novel-coronavirus-2019">https://www.who.int/emergencies/diseases/novel-coronavirus-2019</a>

# 17. APPENDICES

Appendix 1 describes the contraception definitions and requirements applicable for this study.

### **Appendix 1.** Contraception Definitions and Requirements

#### **Definitions (CTFG, 2014)**

Male participants who can father a child with a female partner of childbearing potential must agree to use birth control (2 highly effective methods of contraception including 1 barrier method) during the study period and 90 days after administration of study treatment. Male participants must refrain from donating or banking sperm for 90 days after administration of study treatment. Additionally, female partners of male participants should use highly effective contraception.

A man is considered fertile after puberty unless permanently sterile by bilateral vasectomy with documented aspermia or a bilateral orchiectomy.

### Highly Effective Methods of Contraception

Highly effective methods of contraception are those that have a failure rate of <1% (when implemented consistently and correctly) and include:

- Combined (containing estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (administration may be oral, intravaginal, or transdermal) initiated at least 3 months before the first dose of study treatment; and used in conjunction with a barrier method (e.g., male condom).
- Progestogen-only hormonal contraception associated with inhibition of ovulation (administration may be oral, injectable, or implantable) initiated at least 3 months before the first dose of study treatment; and used in conjunction with a barrier method (e.g., male condom).
- Intrauterine device.
- Intrauterine hormone-releasing system.
- Bilateral tubal ligation
- Vasectomy (provided that the male participant has received medical assessment of surgical success [i.e., azoospermia]).
- Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment[s]); the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant initiated at least 1 month before the first dose of study treatment.

### Acceptable Methods of Contraception That Are Not Considered Highly Effective

Acceptable methods of contraception that result in a failure rate of >1% per year include:

- Progestogen-only hormonal contraception, where inhibition of ovulation is not the primary mode of action.
- Male or female condom with or without spermicide.
- Cap, diaphragm, or sponge with spermicide.
- Double-barrier method (i.e., male condom with either cap, diaphragm, or sponge with spermicide).

### Unacceptable Methods of Contraception

Unacceptable methods of contraception include:

- Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods).
- Withdrawal (i.e., coitus interruptus).
- Spermicides only.
- Lactational amenorrhea.
- Use of female and male condoms together.
- No method at all.
- Cap, diaphragm/sponge without spermicide and without male condom.

# **Appendix 2.** Protocol Amendments

### **Protocol Amendment #1**

Date of Amendment: May 6, 2024

The following updates were made based on regulatory feedback:

| Section | Summary of Change | Justification |
|---|---|---|
| Section 5. | Added injection site reactions and | SAPHRA Recommendation |
| Study | coagulation to safety endpoint, and | |
| Objectives and | specifically mentioned glucose as a | |
| Endpoints | clinical chemistry parameter of interest | |
| Section 8.6.2.1. | Added confirmation that grapefruit juice | SAPHRA Recommendation |
| Meals and | does not impact the metabolism of | |
| Dietary | insulin aspart | |
| Restrictions | | |
| Section 8.6.2.3. | Adjusted prohibition of strenuous | SAPHRA Recommendation |
| Activity | exercise to the entire duration of the | |
| | study | |
| Section 9. | Added Injection Site Assessment to the | SAPHRA Recommendation |
| Study | EOS visit | |
| Procedures | | |
| Section 12. | Updated for consistency with safety | SAPHRA Recommendation |
| Safety | endpoints | |
| Assessments | | |
| Section 12.5. | Provided additional clarity on Injection | SAPHRA Recommendation |
| Injection Site | Site Assessment | |
| Assessment | | |